CLINICAL TRIAL: NCT02612610
Title: A 12-Week Study to Assess the Efficacy and Safety of AF 219 in Subjects With Refractory Chronic Cough
Brief Title: A 12-Week Study in Participants With Refractory Chronic Cough (MK-7264-012)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Afferent Pharmaceuticals, Inc., a subsidiary of Merck & Co., Inc. (Rahway, New Jersey USA) (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 7264-012; AF219-012 (Other: Afferent Pharmaceuticals); 2015-005064-42 (EudraCT Number)
Record Dates: First submitted 2015-11-20; First posted 2015-11-24 (Estimated); Results first posted 2018-02-14 (Actual); Last update posted 2020-06-30 (Actual); Status verified 2020-06

CONDITIONS: Refractory Chronic Cough
MeSH Terms: conditions — Chronic Cough | interventions — Gefapixant

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Placebo (Placebo Comparator): Participants received one matching placebo tablet administered by mouth twice daily for 12 weeks.
  Interventions: Drug: Placebo (for gefapixant)
- Gefapixant 7.5 mg (Experimental): Participants received one 7.5 mg gefapixant tablet administered by mouth twice daily for 12 weeks.
  Interventions: Drug: Gefapixant
- Gefapixant 20 mg (Experimental): Participants received one 20 mg gefapixant tablet administered by mouth twice daily for 12 weeks.
  Interventions: Drug: Gefapixant
- Gefapixant 50 mg (Experimental): Participants received one 50 mg gefapixant tablet administered by mouth twice daily for 12 weeks.
  Interventions: Drug: Gefapixant

INTERVENTIONS:
Drug: Gefapixant — Gefapixant administered as one 7.5 mg, 20 mg, or 50 mg tablet twice daily, depending upon randomization.
  Other Names: AF-219; MK-7264
  Arms: Gefapixant 20 mg; Gefapixant 50 mg; Gefapixant 7.5 mg
Drug: Placebo (for gefapixant)
  Other Names: Dose-matched placebo tablet to gefapixant administered twice daily.
  Arms: Placebo

SUMMARY:
This study is designed to evaluate the efficacy of three dose regimens of gefapixant ([MK-7264] 7.5 mg, 20 mg, and 50 mg) relative to placebo in reducing awake objective cough frequency. The primary hypothesis for this trial is that at least one dose regimen of gefapixant is superior to placebo with respect to the mean change from baseline in awake cough frequency (on the log scale).

ELIGIBILITY:
Inclusion Criteria:

* Women and Men between 18 and 80 years of age inclusive
* Have refractory chronic cough
* Women of child-bearing potential must use 2 forms of acceptable birth control - Have provided written informed consent.
* Are willing and able to comply with all aspects of the protocol

Exclusion Criteria:

* Current smoker
* Forced Expiratory Volume in 1 second (FEV1)/Forced Vital Capacity (FVC) ratio <60%
* History of upper or lower respiratory tract infection or recent significant change in pulmonary status within 4 weeks of the Baseline Visit
* History of opioid use within 1 week of the Baseline Visit
* Body mass index (BMI) <18 kg/m^2 or ≥ 40 kg/m^2
* History of concurrent malignancy or recurrence of malignancy within 2 years prior to Screening (not including subjects with <3 excised basal cell carcinomas)
* Screening systolic blood pressure (SBP) >160 mm Hg or a diastolic blood pressure (DBP) >90 mm Hg
* Clinically significant abnormal electrocardiogram (ECG) at Screening
* Significantly abnormal laboratory tests at Screening
* Pregnant or Breastfeeding
* Other severe, acute, or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with trial participation or investigational product administration or may interfere with the interpretation of trial results and, in the judgment of the Investigator or Sponsor, would make the participant inappropriate for entry into this trial

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 253 (Actual)
Dates: Start 2015-12-15 (Actual); Primary Completion 2016-10-31 (Actual); Study Completion 2016-11-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Afferent Pharmaceuticals Clinical Research, Study Director — Afferent Pharmaceuticals, Inc., a subsidiary of Merck & Co., Inc. (Rahway, New Jersey USA)

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Derived] Schelfhout J, Nguyen AM, Birring SS, Bacci ED, Vernon M, Muccino DR, La Rosa C, Smith JA. Validation and Meaningful Change Thresholds for an Objective Cough Frequency Measurement in Chronic Cough. Lung. 2022 Dec;200(6):717-724. doi: 10.1007/s00408-022-00587-2. Epub 2022 Nov 8. PMID 36348054
- [Derived] Nguyen AM, Schelfhout J, Muccino D, Bacci ED, La Rosa C, Vernon M, Birring SS. Leicester Cough Questionnaire validation and clinically important thresholds for change in refractory or unexplained chronic cough. Ther Adv Respir Dis. 2022 Jan-Dec;16:17534666221099737. doi: 10.1177/17534666221099737. PMID 35614875
- [Derived] Martin Nguyen A, Bacci ED, Vernon M, Birring SS, Rosa C, Muccino D, Schelfhout J. Validation of a visual analog scale for assessing cough severity in patients with chronic cough. Ther Adv Respir Dis. 2021 Jan-Dec;15:17534666211049743. doi: 10.1177/17534666211049743. PMID 34697975
- [Derived] Morice AH, Birring SS, Smith JA, McGarvey LP, Schelfhout J, Martin Nguyen A, Xu ZJ, Wu WC, Muccino DR, Sher MR. Characterization of Patients With Refractory or Unexplained Chronic Cough Participating in a Phase 2 Clinical Trial of the P2X3-Receptor Antagonist Gefapixant. Lung. 2021 Apr;199(2):121-129. doi: 10.1007/s00408-021-00437-7. Epub 2021 Apr 7. PMID 33825965
- [Derived] Smith JA, Kitt MM, Morice AH, Birring SS, McGarvey LP, Sher MR, Li YP, Wu WC, Xu ZJ, Muccino DR, Ford AP; Protocol 012 Investigators. Gefapixant, a P2X3 receptor antagonist, for the treatment of refractory or unexplained chronic cough: a randomised, double-blind, controlled, parallel-group, phase 2b trial. Lancet Respir Med. 2020 Aug;8(8):775-785. doi: 10.1016/S2213-2600(19)30471-0. Epub 2020 Feb 25. PMID 32109425

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of 367 screened, 253 were randomized to treatment with placebo or 7.5 mg, 20 mg, or 50 mg gefapixant. One participant randomized to receive 7.5 mg gefapixant was discontinued before receiving treatment.
Period: Overall Study
Arm/Group | Placebo | Gefapixant 7.5 mg | Gefapixant 20 mg | Gefapixant 50 mg
Started | 63 | 64 | 63 | 63
Treated | 63 | 63 | 63 | 63
Completed | 58 | 56 | 58 | 50
Not Completed | 5 | 8 | 5 | 13
Not completed — Withdrawal by Subject | 1 | 1 | 0 | 2
Not completed — Adverse Event | 2 | 2 | 3 | 10
Not completed — Lost to Follow-up | 0 | 1 | 0 | 0
Not completed — Protocol Violation | 0 | 1 | 1 | 0
Not completed — Lack of Efficacy | 1 | 2 | 0 | 1
Not completed — Physician Decision | 0 | 1 | 0 | 0
Not completed — Noncompliance | 1 | 0 | 0 | 0
Not completed — Cough Improvement | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: All Randomized Participants
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Gefapixant 7.5 mg | Gefapixant 20 mg | Gefapixant 50 mg | Total
Number analyzed (Participants) | 63 | 64 | 63 | 63 | 253
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.0 (10.9) | 59.9 (10.46) | 61.8 (9.13) | 59.3 (9.19) | 60.2 (9.94)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 47 | 48 | 48 | 50 | 193
  Male | 16 | 16 | 15 | 13 | 60

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Awake Objective Cough Frequency After 12 Weeks of Treatment (Day 84)
Description: Awake Objective Cough Frequency (per hour) was defined as the total number of cough events during the monitoring period (in general, 24-hr interval) while the participant was awake divided by the total duration (in hours) for the monitoring period that the participant was awake. 24 hour sound recordings were made at Baseline (Study Day -1) and at Week 12 (Day 84) using a digital recording device. An independent cough monitoring center documented the time of each cough event over the 24 hour period, as well as the time when the participant went to sleep and the time the participant woke. Least-squares (LS) mean change from baseline (in log scale) with associated standard error (SE) reported for each treatment group. Change from Baseline in Awake Objective Cough Frequency = (Post-Treatment Awake Cough Frequency minus Baseline Awake Cough Frequency).
Time Frame: Baseline Visit (Day -1), Day 84
Population: All randomized participants who had taken at least 1 dose of study medication and provided at least 1 baseline and at least one post baseline primary endpoint observation during the treatment period.
Measure: Least Squares Mean (Standard Error); unit: log coughs/hour
Arm/Group | Placebo | Gefapixant 7.5 mg | Gefapixant 20 mg | Gefapixant 50 mg
Number analyzed (Participants) | 61 | 59 | 59 | 57
log coughs/hour | -0.40 (0.11) | -0.64 (0.11) | -0.65 (0.11) | -0.86 (0.11)
Statistical Analysis 1: Comparison: Placebo vs Gefapixant 7.5 mg; Estimated treatment differences (gefapixant vs. placebo) and corresponding 95% confidence intervals (CIs) were estimated using a mixed effect repeated measures (MMRM) model, which included fixed effects for treatment group, visit, country, treatment-by-visit interaction, and Baseline value (on log scale) as a covariate; Test type: Other; p = 0.0971, Mixed Effect Repeated Measures model; LS Mean Difference = -0.25, 95% CI 2-sided [-0.54 to 0.05]
Statistical Analysis 2: Comparison: Placebo vs Gefapixant 20 mg; Estimated treatment differences (gefapixant vs. placebo) and corresponding 95% CIs were estimated using a MMRM model, which included fixed effects for treatment group, visit, country, treatment-by-visit interaction, and Baseline value (on log scale) as a covariate; Test type: Other; p = 0.0928, Mixed Effect Repeated Measures model; LS Mean Difference = -0.25, 95% CI 2-sided [-0.54 to 0.04]
Statistical Analysis 3: Comparison: Placebo vs Gefapixant 50 mg; [analysis description as in outcome 1, analysis 2]; Test type: Other; p = 0.0027, Mixed Effect Repeated Measures model; LS Mean Difference = -0.46, 95% CI 2-sided [-0.76 to -0.16]

2. Secondary Outcome: Change From Baseline in 24-Hour Objective Cough Frequency After 4 Weeks of Treatment (Day 28)
Description: 24-hr Objective Cough Frequency was defined as the total number of cough events during the monitoring period divided by the total duration in hours for the monitoring period (generally 24 hours). 24 hour sound recordings were made at Baseline (Study Day -1) and at Week 4 (Day 28) using a digital recording device. An independent cough monitoring center documented the time of each cough event over the 24 hour period, as well as the time when the participant went to sleep and the time the participant woke. LS mean change from baseline (in log scale) with associated SE reported for each treatment group. Change from Baseline in 24-Hour Objective Cough Frequency = (Post-Treatment 24-Hour Cough Frequency minus Baseline 24-Hour Cough Frequency).
Time Frame: Baseline (Study Day -1), Day 28
Population: All randomized participants who had taken at least 1 dose of study medication and provided at least 1 baseline and at least one post baseline endpoint observation during the treatment period.
Measure: Least Squares Mean (Standard Error); unit: log coughs/hour
Arm/Group | Placebo | Gefapixant 7.5 mg | Gefapixant 20 mg | Gefapixant 50 mg
Number analyzed (Participants) | 61 | 59 | 59 | 57
log coughs/hour | -0.41 (0.10) | -0.59 (0.10) | -0.46 (0.10) | -0.93 (0.10)
Statistical Analysis 1: Comparison: Placebo vs Gefapixant 7.5 mg; Day 28 24-hour Cough Frequency: 7.5 mg gefapixant vs. placebo Day 28 estimated treatment differences (gefapixant vs. placebo) and corresponding 95% CIs were estimated using a MMRM model, which included fixed effects for treatment group, visit, country, treatment-by-visit interaction, and Baseline value (on log scale) as a covariate; Test type: Other; p = 0.1914, Mixed Effect Repeated Measures model; LS Mean Difference = -0.19, 95% CI 2-sided [-0.47 to 0.09]
Statistical Analysis 2: Comparison: Placebo vs Gefapixant 20 mg; Day 28 24-hour Cough Frequency: 20 mg gefapixant vs. placebo Day 28 estimated treatment differences (gefapixant vs. placebo) and corresponding 95% CIs were estimated using a MMRM model, which included fixed effects for treatment group, visit, country, treatment-by-visit interaction, and Baseline value (on log scale) as a covariate; Test type: Other; p = 0.7099, Mixed Effect Repeated Measures model; LS Mean Difference = -0.05, 95% CI 2-sided [-0.33 to 0.23]
Statistical Analysis 3: Comparison: Placebo vs Gefapixant 50 mg; Day 28 24-hour Cough Frequency: 50 mg gefapixant vs. placebo Day 28 estimated treatment differences (gefapixant vs. placebo) and corresponding 95% CIs were estimated using a MMRM model, which included fixed effects for treatment group, visit, country, treatment-by-visit interaction, and Baseline value (on log scale) as a covariate; Test type: Other; p = 0.0003, Mixed Effect Repeated Measures model; LS Mean Difference = -0.52, 95% CI 2-sided [-0.80 to -0.24]

3. Secondary Outcome: Change From Baseline in 24-Hour Objective Cough Frequency After 8 Weeks of Treatment (Day 56)
Description: 24-hr Objective Cough Frequency was defined as the total number of cough events during the monitoring period divided by the total duration in hours for the monitoring period (generally 24 hours). 24 hour sound recordings were made at Baseline (Study Day -1) and at Week 8 (Day 56) using a digital recording device. An independent cough monitoring center documented the time of each cough event over the 24 hour period, as well as the time when the participant went to sleep and the time the participant woke. LS mean change from baseline (in log scale) with associated SE reported for each treatment group. Change from Baseline in 24-Hour Objective Cough Frequency = (Post-Treatment 24-Hour Cough Frequency minus Baseline 24-Hour Cough Frequency).
Time Frame: Baseline (Study Day -1), Day 56
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: log coughs/hour
Arm/Group | Placebo | Gefapixant 7.5 mg | Gefapixant 20 mg | Gefapixant 50 mg
Number analyzed (Participants) | 61 | 59 | 59 | 57
log coughs/hour | -0.31 (0.11) | -0.71 (0.11) | -0.59 (0.11) | -0.93 (0.11)
Statistical Analysis 1: Comparison: Placebo vs Gefapixant 7.5 mg; Day 56 24-hour Cough Frequency: 7.5 mg gefapixant vs. placebo Day 56 estimated treatment differences (gefapixant vs. placebo) and corresponding 95% CIs were estimated using a MMRM model, which included fixed effects for treatment group, visit, country, treatment-by-visit interaction, and Baseline value (on log scale) as a covariate; Test type: Other; p = 0.0099, Mixed Effect Repeated Measures model; LS Mean Difference = -0.40, 95% CI 2-sided [-0.71 to -0.10]
Statistical Analysis 2: Comparison: Placebo vs Gefapixant 20 mg; Day 56 24-hour Cough Frequency: 20 mg gefapixant vs. placebo Day 56 estimated treatment differences (gefapixant vs. placebo) and corresponding 95% CIs were estimated using a MMRM model, which included fixed effects for treatment group, visit, country, treatment-by-visit interaction, and Baseline value (on log scale) as a covariate; Test type: Other; p = 0.0695, Mixed Effect Repeated Measures model; LS Mean Difference = -0.28, 95% CI 2-sided [-0.58 to 0.02]
Statistical Analysis 3: Comparison: Placebo vs Gefapixant 50 mg; Day 56 24-hour Cough Frequency: 50 mg gefapixant vs. placebo Day 56 estimated treatment differences (gefapixant vs. placebo) and corresponding 95% CIs were estimated using a MMRM model, which included fixed effects for treatment group, visit, country, treatment-by-visit interaction, and Baseline value (on log scale) as a covariate; Test type: Other; p = 0.0001, Mixed Effect Repeated Measures model; LS Mean Difference = -0.62, 95% CI 2-sided [-0.93 to -0.31]

4. Secondary Outcome: Change From Baseline in 24-Hour Objective Cough Frequency After 12 Weeks of Treatment (Day 84)
Description: 24-hr Objective Cough Frequency was defined as the total number of cough events during the monitoring period divided by the total duration in hours for the monitoring period (generally 24 hours). 24 hour sound recordings were made at Baseline (Study Day -1) and at Week 12 (Day 84) using a digital recording device. An independent cough monitoring center documented the time of each cough event over the 24 hour period, as well as the time when the participant went to sleep and the time the participant woke. LS mean change from baseline (in log scale) with associated SE reported for each treatment group. Change from Baseline in 24-Hour Objective Cough Frequency = (Post-Treatment 24-Hour Cough Frequency minus Baseline 24-Hour Cough Frequency).
Time Frame: Baseline (Study Day -1), Day 84
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: log coughs/hour
Arm/Group | Placebo | Gefapixant 7.5 mg | Gefapixant 20 mg | Gefapixant 50 mg
Number analyzed (Participants) | 61 | 59 | 59 | 57
log coughs/hour | -0.39 (0.10) | -0.62 (0.10) | -0.64 (0.10) | -0.86 (0.11)
Statistical Analysis 1: Comparison: Placebo vs Gefapixant 7.5 mg; Day 84 24-hour Cough Frequency: 7.5 mg gefapixant vs. placebo Day 84 estimated treatment differences (gefapixant vs. placebo) and corresponding 95% CIs were estimated using a MMRM model, which included fixed effects for treatment group, visit, country, treatment-by-visit interaction, and Baseline value (on log scale) as a covariate; Test type: Other; p = 0.0991, Mixed Effect Repeated Measures model; LS Mean Difference = -0.24, 95% CI 2-sided [-0.52 to 0.04]
Statistical Analysis 2: Comparison: Placebo vs Gefapixant 20 mg; Day 84 24-hour Cough Frequency: 20 mg gefapixant vs. placebo Day 84 estimated treatment differences (gefapixant vs. placebo) and corresponding 95% CIs were estimated using a MMRM model, which included fixed effects for treatment group, visit, country, treatment-by-visit interaction, and Baseline value (on log scale) as a covariate; Test type: Other; p = 0.0811, Mixed Effect Repeated Measures model; LS Mean Difference = -0.25, 95% CI 2-sided [-0.53 to 0.03]
Statistical Analysis 3: Comparison: Placebo vs Gefapixant 50 mg; Day 84 24-hour Cough Frequency: 50 mg gefapixant vs. placebo Day 84 estimated treatment differences (gefapixant vs. placebo) and corresponding 95% CIs were estimated using a MMRM model, which included fixed effects for treatment group, visit, country, treatment-by-visit interaction, and Baseline value (on log scale) as a covariate; Test type: Other; p = 0.0014, Mixed Effect Repeated Measures model; LS Mean Difference = -0.47, 95% CI 2-sided [-0.76 to -0.19]

5. Secondary Outcome: Change From Baseline in Awake Objective Cough Frequency After 4 Weeks of Treatment (Day 28)
Description: Awake Objective Cough Frequency (per hour) was defined as the total number of cough events during the monitoring period (in general, 24-hr interval) while the participant was awake divided by the total duration (in hours) for the monitoring period that the participant was awake. 24 hour sound recordings were made at Baseline (Study Day -1) and at Week 4 (Day 28) using a digital recording device. An independent cough monitoring center documented the time of each cough event over the 24 hour period, as well as the time when the participant went to sleep and the time the participant woke. LS mean change from baseline (in log scale) with associated SE reported for each treatment group. Change from Baseline in Awake Objective Cough Frequency = (Post-Treatment Awake Cough Frequency minus Baseline Awake Cough Frequency).
Time Frame: Baseline (Study Day -1), Day 28,
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: log coughs/hour
Arm/Group | Placebo | Gefapixant 7.5 mg | Gefapixant 20 mg | Gefapixant 50 mg
Number analyzed (Participants) | 61 | 59 | 59 | 57
log coughs/hour | -0.41 (0.10) | -0.62 (0.10) | -0.48 (0.10) | -0.90 (0.11)
Statistical Analysis 1: Comparison: Placebo vs Gefapixant 7.5 mg; Day 28 Awake Cough Frequency: 7.5 mg gefapixant vs. placebo Day 28 estimated treatment differences (gefapixant vs. placebo) and corresponding 95% CIs were estimated using a MMRM model, which included fixed effects for treatment group, visit, country, treatment-by-visit interaction, and Baseline value (on log scale) as a covariate; Test type: Other; p = 0.1468, Mixed Effect Repeated Measures model; LS Mean Difference = -0.21, 95% CI 2-sided [-0.50 to 0.07]
Statistical Analysis 2: Comparison: Placebo vs Gefapixant 20 mg; Day 28 Awake Cough Frequency: 20 mg gefapixant vs. placebo Day 28 estimated treatment differences (gefapixant vs. placebo) and corresponding 95% CIs were estimated using a MMRM model, which included fixed effects for treatment group, visit, country, treatment-by-visit interaction, and Baseline value (on log scale) as a covariate; Test type: Other; p = 0.5874, Mixed Effect Repeated Measures model; LS Mean Difference = -0.08, 95% CI 2-sided [-0.36 to 0.20]
Statistical Analysis 3: Comparison: Placebo vs Gefapixant 50 mg; [analysis description as in outcome 2, analysis 3]; Test type: Other; p = 0.0008, Mixed Effect Repeated Measures model; LS Mean Difference = -0.49, 95% CI 2-sided [-0.78 to -0.21]

6. Secondary Outcome: Change From Baseline in Awake Objective Cough Frequency After 8 Weeks of Treatment (Day 56)
Description: Awake Objective Cough Frequency (per hour) was defined as the total number of cough events during the monitoring period (in general, 24-hr interval) while the participant was awake divided by the total duration (in hours) for the monitoring period that the participant was awake. 24 hour sound recordings were made at Baseline (Study Day -1) and at Week 8 (Day 56) using a digital recording device. An independent cough monitoring center documented the time of each cough event over the 24 hour period, as well as the time when the participant went to sleep and the time the participant woke. LS mean change from baseline (in log scale) with associated SE reported for each treatment group. Change from Baseline in Awake Objective Cough Frequency = (Post-Treatment Awake Cough Frequency minus Baseline Awake Cough Frequency).
Time Frame: Baseline (Study Day -1), Day 56
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: log coughs/hour
Arm/Group | Placebo | Gefapixant 7.5 mg | Gefapixant 20 mg | Gefapixant 50 mg
Number analyzed (Participants) | 61 | 59 | 59 | 57
log coughs/hour | -0.31 (0.11) | -0.70 (0.12) | -0.63 (0.11) | -0.90 (0.12)
Statistical Analysis 1: Comparison: Placebo vs Gefapixant 7.5 mg; Day 56 Awake Cough Frequency: 7.5 mg gefapixant vs. placebo Day 56 estimated treatment differences (gefapixant vs. placebo) and corresponding 95% CIs were estimated using a MMRM model, which included fixed effects for treatment group, visit, country, treatment-by-visit interaction, and Baseline value (on log scale) as a covariate; Test type: Other; p = 0.0177, Mixed Effect Repeated Measures model; Mixed Effect Repeated Measures model = -0.39, 95% CI 2-sided [-0.70 to -0.07]
Statistical Analysis 2: Comparison: Placebo vs Gefapixant 20 mg; Day 56 Awake Cough Frequency: 20 mg gefapixant vs. placebo Day 56 estimated treatment differences (gefapixant vs. placebo) and corresponding 95% CIs were estimated using a MMRM model, which included fixed effects for treatment group, visit, country, treatment-by-visit interaction, and Baseline value (on log scale) as a covariate; Test type: Other; p = 0.0498, Mixed Effect Repeated Measures model; LS Mean Difference = -0.32, 95% CI 2-sided [-0.63 to -0.00]
Statistical Analysis 3: Comparison: Placebo vs Gefapixant 50 mg; Day 56 Awake Cough Frequency: 50 mg gefapixant vs. placebo Day 56 estimated treatment differences (gefapixant vs. placebo) and corresponding 95% CIs were estimated using a MMRM model, which included fixed effects for treatment group, visit, country, treatment-by-visit interaction, and Baseline value (on log scale) as a covariate; Test type: Other; p = 0.0004, Mixed Effect Repeated Measures model; LS Mean Difference = -0.59, 95% CI 2-sided [-0.92 to -0.27]

7. Secondary Outcome: Change From Baseline in Awake Objective Cough Frequency at the Follow-up Visit (Day 98)
Description: Awake Objective Cough Frequency (per hour) was defined as the total number of cough events during the monitoring period (in general, 24-hr interval) while the participant was awake divided by the total duration (in hours) for the monitoring period that the participant was awake. 24 hour sound recordings were made at Baseline (Study Day -1) and at the Follow-up visit (Day 98) using a digital recording device. An independent cough monitoring center documented the time of each cough event over the 24 hour period, as well as the time when the participant went to sleep and the time the participant woke. Change from Baseline in Awake Objective Cough Frequency = (Post-Treatment Awake Cough Frequency minus Baseline Awake Cough Frequency).
Time Frame: Baseline (Study Day -1), Day 98
Population: All randomized participants who had taken at least 1 dose of study medication and provided baseline and follow-up visit (Day 98) data during the treatment period.
Measure: Mean (Standard Deviation); unit: coughs/hour
Arm/Group | Placebo | Gefapixant 7.5 mg | Gefapixant 20 mg | Gefapixant 50 mg
Number analyzed (Participants) | 58 | 55 | 56 | 51
coughs/hour | -6.4 (22.72) | -9.3 (47.72) | -7.4 (29.24) | -16.2 (39.00)

8. Secondary Outcome: Change From Baseline in Cough Severity Visual Analogue Scale (VAS) After 4 Weeks of Treatment (Day 28)
Description: Cough VAS was scored from 0 to 100 using a 100 mm visual analogue scale. Participants were asked to mark on a 100 mm scale between 0 (no cough) and 100 (the worst cough severity). Cough VAS was evaluated at Baseline (Study Day -1) and at Week 4 (Day 28). Baseline cough VAS was defined as the cough VAS at Baseline (Study Day -1). LS mean change from baseline with associated SE reported for each treatment group.
Time Frame: Baseline (Study Day -1), Day 28
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Gefapixant 7.5 mg | Gefapixant 20 mg | Gefapixant 50 mg
Number analyzed (Participants) | 61 | 59 | 59 | 57
units on a scale | -15.2 (3.02) | -21.6 (3.05) | -18.1 (3.04) | -25. (3.09)
Statistical Analysis 1: Comparison: Placebo vs Gefapixant 7.5 mg; Day 28 Cough Severity VAS: 7.5 mg gefapixant vs. placebo Day 28 estimated treatment differences (gefapixant vs. placebo) and corresponding 95% CIs were estimated using a MMRM model, which included fixed effects for treatment group, visit, country, treatment-by-visit interaction, and Baseline value as a covariate; Test type: Other; p = 0.1318, Mixed Effect Repeated Measures model; LS Mean Difference = -6.4, 95% CI 2-sided [-14.8 to 1.9]
Statistical Analysis 2: Comparison: Placebo vs Gefapixant 20 mg; Day 28 Cough Severity VAS: 20 mg gefapixant vs. placebo Day 28 estimated treatment differences (gefapixant vs. placebo) and corresponding 95% CIs were estimated using a MMRM model, which included fixed effects for treatment group, visit, country, treatment-by-visit interaction, and Baseline value as a covariate; Test type: Other; p = 0.4917, Mixed Effect Repeated Measures model; LS Mean Difference = -2.9, 95% CI 2-sided [-11.3 to 5.4]
Statistical Analysis 3: Comparison: Placebo vs Gefapixant 50 mg; Day 28 Cough Severity VAS: 50 mg gefapixant vs. placebo Day 28 estimated treatment differences (gefapixant vs. placebo) and corresponding 95% CIs were estimated using a MMRM model, which included fixed effects for treatment group, visit, country, treatment-by-visit interaction, and Baseline value as a covariate; Test type: Other; p = 0.0228, Mixed Effect Repeated Measures model; LS Mean Difference = -9.8, 95% CI 2-sided [-18.2 to -1.4]

9. Secondary Outcome: Change From Baseline in Cough Severity VAS After 8 Weeks of Treatment (Day 56)
Description: Cough VAS was scored from 0 to 100 using a 100 mm visual analogue scale. Participants were asked to mark on a 100 mm scale between 0 (no cough) and 100 (the worst cough severity). Cough VAS was evaluated at Baseline (Study Day -1) and at Week 8 (Day 56). Baseline cough VAS was defined as the cough VAS at Baseline (Study Day -1). LS mean change from baseline with associated SE reported for each treatment group.
Time Frame: Baseline (Study Day -1), Day 56
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Gefapixant 7.5 mg | Gefapixant 20 mg | Gefapixant 50 mg
Number analyzed (Participants) | 61 | 59 | 59 | 57
units on a scale | -16.1 (3.18) | -18.8 (3.19) | -19.4 (3.18) | -26.9 (3.33)
Statistical Analysis 1: Comparison: Placebo vs Gefapixant 7.5 mg; Day 56 Cough Severity VAS: 7.5 mg gefapixant vs. placebo Day 56 estimated treatment differences (gefapixant vs. placebo) and corresponding 95% CIs were estimated using a MMRM model, which included fixed effects for treatment group, visit, country, treatment-by-visit interaction, and Baseline value as a covariate; Test type: Other; p = 0.5540, Mixed Effect Repeated Measures model; LS Mean Difference = -2.6, 95% CI 2-sided [-11.5 to 6.2]
Statistical Analysis 2: Comparison: Placebo vs Gefapixant 20 mg; Day 56 Cough Severity VAS: 20 mg gefapixant vs. placebo Day 56 estimated treatment differences (gefapixant vs. placebo) and corresponding 95% CIs were estimated using a MMRM model, which included fixed effects for treatment group, visit, country, treatment-by-visit interaction, and Baseline value as a covariate; Test type: Other; p = 0.4702, Mixed Effect Repeated Measures model; LS Mean Difference = -3.2, 95% CI 2-sided [-12.0 to 5.6]
Statistical Analysis 3: Comparison: Placebo vs Gefapixant 50 mg; Day 56 Cough Severity VAS: 50 mg gefapixant vs. placebo Day 56 estimated treatment differences (gefapixant vs. placebo) and corresponding 95% CIs were estimated using a MMRM model, which included fixed effects for treatment group, visit, country, treatment-by-visit interaction, and Baseline value as a covariate; Test type: Other; p = 0.0197, Mixed Effect Repeated Measures model; LS Mean Difference = -10.7, 95% CI 2-sided [-19.8 to -1.7]

10. Secondary Outcome: Change From Baseline in Cough Severity VAS After 12 Weeks of Treatment (Day 84)
Description: Cough VAS was scored from 0 to 100 using a 100 mm visual analogue scale. Participants were asked to mark on a 100 mm scale between 0 (no cough) and 100 (the worst cough severity). Cough VAS was evaluated at Baseline (Study Day -1) and at Week 12 (Day 84). Baseline cough VAS was defined as the cough VAS at Baseline (Study Day -1). LS mean change from baseline with associated SE reported for each treatment group.
Time Frame: Baseline (Study Day -1), Day 84
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Gefapixant 7.5 mg | Gefapixant 20 mg | Gefapixant 50 mg
Number analyzed (Participants) | 61 | 59 | 59 | 57
units on a scale | -16.7 (3.04) | -21.1 (3.08) | -23.1 (3.05) | -27.9 (3.16)
Statistical Analysis 1: Comparison: Placebo vs Gefapixant 7.5 mg; Day 84 Cough Severity VAS: 7.5 mg gefapixant vs. placebo Day 84 estimated treatment differences (gefapixant vs. placebo) and corresponding 95% CIs were estimated using a MMRM model, which included fixed effects for treatment group, visit, country, treatment-by-visit interaction, and Baseline value as a covariate; Test type: Other; p = 0.3020, Mixed Effect Repeated Measures model; LS Mean Difference = -4.4, 95% CI 2-sided [-12.9 to 4.0]
Statistical Analysis 2: Comparison: Placebo vs Gefapixant 20 mg; Day 84 Cough Severity VAS: 20 mg gefapixant vs. placebo Day 84 estimated treatment differences (gefapixant vs. placebo) and corresponding 95% CIs were estimated using a MMRM model, which included fixed effects for treatment group, visit, country, treatment-by-visit interaction, and Baseline value as a covariate; Test type: Other; p = 0.1365, Mixed Effect Repeated Measures model; LS Mean Difference = -6.4, 95% CI 2-sided [-14.8 to 2.0]
Statistical Analysis 3: Comparison: Placebo vs Gefapixant 50 mg; Day 84 Cough Severity VAS: 50 mg gefapixant vs. placebo Day 84 estimated treatment differences (gefapixant vs. placebo) and corresponding 95% CIs were estimated using a MMRM model, which included fixed effects for treatment group, visit, country, treatment-by-visit interaction, and Baseline value as a covariate; Test type: Other; p = 0.0108, Mixed Effect Repeated Measures model; LS Mean Difference = -11.2, 95% CI 2-sided [-19.7 to -2.6]

11. Secondary Outcome: Change From Baseline in Cough Severity VAS At Day 85/Early Termination
Description: Cough VAS was scored from 0 to 100 using a 100 mm visual analogue scale. Participants were asked to mark on a 100 mm scale between 0 (no cough) and 100 (the worst cough severity). Cough VAS was evaluated at Baseline (Study Day -1) and at Day 85/Early Termination. Baseline cough VAS was defined as the cough VAS at Baseline (Study Day -1). LS mean change from baseline with associated SE reported for each treatment group.
Time Frame: Baseline (Study Day -1), Day 85
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Gefapixant 7.5 mg | Gefapixant 20 mg | Gefapixant 50 mg
Number analyzed (Participants) | 61 | 59 | 59 | 57
units on a scale | -15.2 (3.00) | -19.2 (3.04) | -23.4 (3.03) | -31.1 (3.09)
Statistical Analysis 1: Comparison: Placebo vs Gefapixant 7.5 mg; Day 85/Early Termination Cough Severity VAS: 7.5 mg gefapixant vs. placebo Day 85/Early Termination estimated treatment differences (gefapixant vs. placebo) and corresponding 95% CIs were estimated using a MMRM model, which included fixed effects for treatment group, visit, country, treatment-by-visit interaction, and Baseline value as a covariate; Test type: Other; p = 0.3509, Mixed Effect Repeated Measures model; LS Mean Difference = -4.0, 95% CI 2-sided [-12.3 to 4.4]
Statistical Analysis 2: Comparison: Placebo vs Gefapixant 20 mg; [analysis description as in outcome 11, analysis 1]; Test type: Other; p = 0.0519, Mixed Effect Repeated Measures model; LS Mean Difference = -8.2, 95% CI 2-sided [-16.6 to 0.1]
Statistical Analysis 3: Comparison: Placebo vs Gefapixant 50 mg; Day 85/Early Termination Cough Severity VAS: 50 mg gefapixant vs. placebo Day 85/Early Termination estimated treatment differences (gefapixant vs. placebo) and corresponding 95% CIs were estimated using a MMRM model, which included fixed effects for treatment group, visit, country, treatment-by-visit interaction, and Baseline value as a covariate; Test type: Other; p = 0.0003, Mixed Effect Repeated Measures model; LS Mean Difference = -15.9, 95% CI 2-sided [-24.3 to -7.5]

12. Secondary Outcome: Percentage of Participants With ≥70%, ≥50%, and ≥30% Change From Baseline in Awake Objective Cough Frequency After 4 Weeks of Treatment (Day 28)
Description: Awake Objective Cough Frequency (per hour) was defined as the total number of cough events during the monitoring period (in general, 24-hr interval) while the participant was awake divided by the total duration (in hours) for the monitoring period that the participant was awake. 24 hour sound recordings were made at Baseline (Study Day -1) and at Week 4 (Day 28) using a digital recording device. An independent cough monitoring center documented the time of each cough event over the 24 hour period, as well as the time when the participant went to sleep and the time the participant woke. The percentage of participants that met responder criteria for ≥70%, ≥50%, and ≥30% change (reduction) from baseline levels in Awake Objective Cough Frequency were reported for each treatment group at Day 28.
Time Frame: Baseline (Study Day -1), Day 28
Population: All randomized participants who had taken at least 1 dose of study medication and provided at least 1 baseline and at least one Day 28 endpoint observation during the treatment period.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Gefapixant 7.5 mg | Gefapixant 20 mg | Gefapixant 50 mg
Number analyzed (Participants) | 60 | 55 | 59 | 55
percentage of participants
  ≥70% Change | 15.0 (0.10) | 25.5 (0.10) | 16.9 (0.10) | 34.5 (0.10)
  ≥50% Change | 23.3 (0.11) | 38.2 (0.11) | 30.5 (0.11) | 47.3 (0.11)
  ≥30% Change | 46.7 (0.10) | 63.6 (0.10) | 50.8 (0.10) | 60.0 (0.11)
Statistical Analysis 1: Comparison: Placebo vs Gefapixant 7.5 mg; Day 28: ≥70% Change: 7.5 mg gefapixant vs. placebo Cough frequency responder endpoints were analyzed by a generalized linear mixed model (GLMM) with treatment, visit, and treatment by visit interaction, and country as fixed effects. Comparison of response rates between each gefapixant treatment group and placebo was conducted using the stratified Cochran Mantel Haenszel (CMH) test (stratified by country, unless stated otherwise). Missing data was categorized as discontinued or missing; Test type: Superiority or Other; p = 0.1387, Cochran-Mantel-Haenszel
Statistical Analysis 2: Comparison: Placebo vs Gefapixant 20 mg; Day 28: ≥70% Change: 20 mg gefapixant vs. placebo Cough frequency responder endpoints were analyzed by a GLMM with treatment, visit, and treatment by visit interaction, and country as fixed effects. Comparison of response rates between each gefapixant treatment group and placebo was conducted using the stratified CMH test (stratified by country, unless stated otherwise). Missing data was categorized as discontinued or missing; Test type: Superiority or Other; p = 0.7238, Cochran-Mantel-Haenszel
Statistical Analysis 3: Comparison: Placebo vs Gefapixant 50 mg; Day 28: ≥70% Change: 50 mg gefapixant vs. placebo Cough frequency responder endpoints were analyzed by a GLMM with treatment, visit, and treatment by visit interaction, and country as fixed effects. Comparison of response rates between each gefapixant treatment group and placebo was conducted using the stratified CMH test (stratified by country, unless stated otherwise). Missing data was categorized as discontinued or missing; Test type: Superiority or Other; p = 0.0144, Cochran-Mantel-Haenszel
Statistical Analysis 4: Comparison: Placebo vs Gefapixant 7.5 mg; Day 28: ≥50% Change: 7.5 mg gefapixant vs. placebo Cough frequency responder endpoints were analyzed by a GLMM with treatment, visit, and treatment by visit interaction, and country as fixed effects. Comparison of response rates between each gefapixant treatment group and placebo was conducted using the stratified CMH test (stratified by country, unless stated otherwise). Missing data was categorized as discontinued or missing; Test type: Superiority or Other; p = 0.0922, Cochran-Mantel-Haenszel
Statistical Analysis 5: Comparison: Placebo vs Gefapixant 20 mg; Day 28: ≥50% Change: 20 mg gefapixant vs. placebo Cough frequency responder endpoints were analyzed by a GLMM with treatment, visit, and treatment by visit interaction, and country as fixed effects. Comparison of response rates between each gefapixant treatment group and placebo was conducted using the stratified CMH test (stratified by country, unless stated otherwise). Missing data was categorized as discontinued or missing; Test type: Superiority or Other; p = 0.3812, Cochran-Mantel-Haenszel
Statistical Analysis 6: Comparison: Placebo vs Gefapixant 50 mg; Day 28: ≥50% Change: 50 mg gefapixant vs. placebo Cough frequency responder endpoints were analyzed by a GLMM with treatment, visit, and treatment by visit interaction, and country as fixed effects. Comparison of response rates between each gefapixant treatment group and placebo was conducted using the stratified CMH test (stratified by country, unless stated otherwise). Missing data was categorized as discontinued or missing; Test type: Superiority or Other; p = 0.0088, Cochran-Mantel-Haenszel
Statistical Analysis 7: Comparison: Placebo vs Gefapixant 7.5 mg; Day 28: ≥30% Change: 7.5 mg gefapixant vs. placebo Cough frequency responder endpoints were analyzed by a GLMM with treatment, visit, and treatment by visit interaction, and country as fixed effects. Comparison of response rates between each gefapixant treatment group and placebo was conducted using the stratified CMH test (stratified by country, unless stated otherwise). Missing data was categorized as discontinued or missing; Test type: Superiority or Other; p = 0.0653, Cochran-Mantel-Haenszel
Statistical Analysis 8: Comparison: Placebo vs Gefapixant 20 mg; Day 28: ≥30% Change: 20 mg gefapixant vs. placebo Cough frequency responder endpoints were analyzed by a GLMM with treatment, visit, and treatment by visit interaction, and country as fixed effects. Comparison of response rates between each gefapixant treatment group and placebo was conducted using the stratified CMH test (stratified by country, unless stated otherwise). Missing data was categorized as discontinued or missing; Test type: Superiority or Other; p = 0.6443, Cochran-Mantel-Haenszel
Statistical Analysis 9: Comparison: Placebo vs Gefapixant 50 mg; Day 28: ≥30% Change: 50 mg gefapixant vs. placebo Cough frequency responder endpoints were analyzed by a GLMM with treatment, visit, and treatment by visit interaction, and country as fixed effects. Comparison of response rates between each gefapixant treatment group and placebo was conducted using the stratified CMH test (stratified by country, unless stated otherwise). Missing data was categorized as discontinued or missing; Test type: Superiority or Other; p = 0.1511, Cochran-Mantel-Haenszel

13. Secondary Outcome: Percentage of Participants With ≥70%, ≥50%, and ≥30% Change From Baseline in Awake Objective Cough Frequency After 8 Weeks of Treatment (Day 56)
Description: Awake Objective Cough Frequency (per hour) was defined as the total number of cough events during the monitoring period (in general, 24-hr interval) while the participant was awake divided by the total duration (in hours) for the monitoring period that the participant was awake. 24 hour sound recordings were made at Baseline (Study Day -1) and at Week 8 (Day 56) using a digital recording device. An independent cough monitoring center documented the time of each cough event over the 24 hour period, as well as the time when the participant went to sleep and the time the participant woke. The percentage of participants that met responder criteria for ≥70%, ≥50%, and ≥30% change (reduction) from baseline levels in Awake Objective Cough Frequency were reported for each treatment group at Day 56.
Time Frame: Baseline (Study Day -1), Day 56
Population: All randomized participants who had taken at least 1 dose of study medication and provided at least 1 baseline and at least one Day 56 endpoint observation during the treatment period.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Gefapixant 7.5 mg | Gefapixant 20 mg | Gefapixant 50 mg
Number analyzed (Participants) | 57 | 56 | 59 | 51
percentage of participants
  ≥70% Change | 10.5 (0.10) | 32.1 (0.10) | 22.0 (0.10) | 31.4 (0.10)
  ≥50% Change | 26.3 (0.11) | 46.4 (0.11) | 39.0 (0.11) | 54.9 (0.11)
  ≥30% Change | 47.4 (0.10) | 64.3 (0.10) | 55.9 (0.10) | 72.5 (0.11)
Statistical Analysis 1: Comparison: Placebo vs Gefapixant 7.5 mg; Day 56: ≥70% Change: 7.5 mg gefapixant vs. placebo Cough frequency responder endpoints were analyzed by a generalized linear mixed model (GLMM) with treatment, visit, and treatment by visit interaction, and country as fixed effects. Comparison of response rates between each gefapixant treatment group and placebo was conducted using the stratified Cochran Mantel Haenszel (CMH) test (stratified by country, unless stated otherwise). Missing data was categorized as discontinued or missing; Test type: Superiority or Other; p = 0.0045, Cochran-Mantel-Haenszel
Statistical Analysis 2: Comparison: Placebo vs Gefapixant 20 mg; Day 56: ≥70% Change: 20 mg gefapixant vs. placebo Cough frequency responder endpoints were analyzed by a GLMM with treatment, visit, and treatment by visit interaction, and country as fixed effects. Comparison of response rates between each gefapixant treatment group and placebo was conducted using the stratified CMH test (stratified by country, unless stated otherwise). Missing data was categorized as discontinued or missing; Test type: Superiority or Other; p = 0.0947, Cochran-Mantel-Haenszel
Statistical Analysis 3: Comparison: Placebo vs Gefapixant 50 mg; Day 56: ≥70% Change: 50 mg gefapixant vs. placebo Cough frequency responder endpoints were analyzed by a GLMM with treatment, visit, and treatment by visit interaction, and country as fixed effects. Comparison of response rates between each gefapixant treatment group and placebo was conducted using the stratified CMH test (stratified by country, unless stated otherwise). Missing data was categorized as discontinued or missing; Test type: Superiority or Other; p = 0.0080, Cochran-Mantel-Haenszel
Statistical Analysis 4: Comparison: Placebo vs Gefapixant 7.5 mg; Day 56: ≥50% Change: 7.5 mg gefapixant vs. placebo Cough frequency responder endpoints were analyzed by a GLMM with treatment, visit, and treatment by visit interaction, and country as fixed effects. Comparison of response rates between each gefapixant treatment group and placebo was conducted using the stratified CMH test (stratified by country, unless stated otherwise). Missing data was categorized as discontinued or missing; Test type: Superiority or Other; p = 0.0283, Cochran-Mantel-Haenszel
Statistical Analysis 5: Comparison: Placebo vs Gefapixant 20 mg; Day 56: ≥50% Change: 20 mg gefapixant vs. placebo Cough frequency responder endpoints were analyzed by a GLMM with treatment, visit, and treatment by visit interaction, and country as fixed effects. Comparison of response rates between each gefapixant treatment group and placebo was conducted using the stratified CMH test (stratified by country, unless stated otherwise). Missing data was categorized as discontinued or missing; Test type: Superiority or Other; p = 0.1493, Cochran-Mantel-Haenszel
Statistical Analysis 6: Comparison: Placebo vs Gefapixant 50 mg; Day 56: ≥50% Change: 50 mg gefapixant vs. placebo Cough frequency responder endpoints were analyzed by a GLMM with treatment, visit, and treatment by visit interaction, and country as fixed effects. Comparison of response rates between each gefapixant treatment group and placebo was conducted using the stratified CMH test (stratified by country, unless stated otherwise). Missing data was categorized as discontinued or missing; Test type: Superiority or Other; p = 0.0026, Cochran-Mantel-Haenszel
Statistical Analysis 7: Comparison: Placebo vs Gefapixant 7.5 mg; Day 56: ≥30% Change: 7.5 mg gefapixant vs. placebo Cough frequency responder endpoints were analyzed by a GLMM with treatment, visit, and treatment by visit interaction, and country as fixed effects. Comparison of response rates between each gefapixant treatment group and placebo was conducted using the stratified CMH test (stratified by country, unless stated otherwise). Missing data was categorized as discontinued or missing; Test type: Superiority or Other; p = 0.0652, Cochran-Mantel-Haenszel
Statistical Analysis 8: Comparison: Placebo vs Gefapixant 20 mg; Day 56: ≥30% Change: 20 mg gefapixant vs. placebo Cough frequency responder endpoints were analyzed by a GLMM with treatment, visit, and treatment by visit interaction, and country as fixed effects. Comparison of response rates between each gefapixant treatment group and placebo was conducted using the stratified CMH test (stratified by country, unless stated otherwise). Missing data was categorized as discontinued or missing; Test type: Superiority or Other; p = 0.3601, Cochran-Mantel-Haenszel
Statistical Analysis 9: Comparison: Placebo vs Gefapixant 50 mg; Day 56: ≥30% Change: 50 mg gefapixant vs. placebo Cough frequency responder endpoints were analyzed by a GLMM with treatment, visit, and treatment by visit interaction, and country as fixed effects. Comparison of response rates between each gefapixant treatment group and placebo was conducted using the stratified CMH test (stratified by country, unless stated otherwise). Missing data was categorized as discontinued or missing; Test type: Superiority or Other; p = 0.0086, Cochran-Mantel-Haenszel

14. Secondary Outcome: Percentage of Participants With ≥70%, ≥50%, and ≥30% Change From Baseline in Awake Objective Cough Frequency After 12 Weeks of Treatment (Day 84)
Description: Awake Objective Cough Frequency (per hour) was defined as the total number of cough events during the monitoring period (in general, 24-hr interval) while the participant was awake divided by the total duration (in hours) for the monitoring period that the participant was awake. 24 hour sound recordings were made at Baseline (Study Day -1) and at Week 12 (Day 84) using a digital recording device. An independent cough monitoring center documented the time of each cough event over the 24 hour period, as well as the time when the participant went to sleep and the time the participant woke. The percentage of participants that met responder criteria for ≥70%, ≥50%, and ≥30% change (reduction) from baseline levels in Awake Objective Cough Frequency were reported for each treatment group at Day 84.
Time Frame: Baseline (Study Day -1), Day 84
Population: All randomized participants who had taken at least 1 dose of study medication and provided at least 1 baseline and at least one Day 84 endpoint observation during the treatment period.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Gefapixant 7.5 mg | Gefapixant 20 mg | Gefapixant 50 mg
Number analyzed (Participants) | 57 | 56 | 56 | 51
percentage of participants
  ≥70% Change | 15.8 (0.10) | 21.4 (0.10) | 23.2 (0.10) | 31.4 (0.10)
  ≥50% Change | 24.6 (0.11) | 44.6 (0.11) | 32.1 (0.11) | 51.0 (0.11)
  ≥30% Change | 43.9 (0.10) | 64.3 (0.10) | 48.2 (0.10) | 80.4 (0.11)
Statistical Analysis 1: Comparison: Placebo vs Gefapixant 7.5 mg; Day 84: ≥70% Change: 7.5 mg gefapixant vs. placebo Cough frequency responder endpoints were analyzed by a generalized linear mixed model (GLMM) with treatment, visit, and treatment by visit interaction, and country as fixed effects. Comparison of response rates between each gefapixant treatment group and placebo was conducted using the stratified Cochran Mantel Haenszel (CMH) test (stratified by country, unless stated otherwise). Missing data was categorized as discontinued or missing; Test type: Superiority or Other; p = 0.3893, Cochran-Mantel-Haenszel
Statistical Analysis 2: Comparison: Placebo vs Gefapixant 20 mg; Day 84: ≥70% Change: 20 mg gefapixant vs. placebo Cough frequency responder endpoints were analyzed by a GLMM with treatment, visit, and treatment by visit interaction, and country as fixed effects. Comparison of response rates between each gefapixant treatment group and placebo was conducted using the stratified CMH test (stratified by country, unless stated otherwise). Missing data was categorized as discontinued or missing; Test type: Superiority or Other; p = 0.2803, Cochran-Mantel-Haenszel
Statistical Analysis 3: Comparison: Placebo vs Gefapixant 50 mg; Day 84: ≥70% Change: 50 mg gefapixant vs. placebo Cough frequency responder endpoints were analyzed by a GLMM with treatment, visit, and treatment by visit interaction, and country as fixed effects. Comparison of response rates between each gefapixant treatment group and placebo was conducted using the stratified CMH test (stratified by country, unless stated otherwise). Missing data was categorized as discontinued or missing; Test type: Superiority or Other; p = 0.0427, Cochran-Mantel-Haenszel
Statistical Analysis 4: Comparison: Placebo vs Gefapixant 7.5 mg; Day 84: ≥50% Change: 7.5 mg gefapixant vs. placebo Cough frequency responder endpoints were analyzed by a GLMM with treatment, visit, and treatment by visit interaction, and country as fixed effects. Comparison of response rates between each gefapixant treatment group and placebo was conducted using the stratified CMH test (stratified by country, unless stated otherwise). Missing data was categorized as discontinued or missing; Test type: Superiority or Other; p = 0.0209, Cochran-Mantel-Haenszel
Statistical Analysis 5: Comparison: Placebo vs Gefapixant 20 mg; Day 84: ≥50% Change: 20 mg gefapixant vs. placebo Cough frequency responder endpoints were analyzed by a GLMM with treatment, visit, and treatment by visit interaction, and country as fixed effects. Comparison of response rates between each gefapixant treatment group and placebo was conducted using the stratified CMH test (stratified by country, unless stated otherwise). Missing data was categorized as discontinued or missing; Test type: Superiority or Other; p = 0.3401, Cochran-Mantel-Haenszel
Statistical Analysis 6: Comparison: Placebo vs Gefapixant 50 mg; Day 84: ≥50% Change: 50 mg gefapixant vs. placebo Cough frequency responder endpoints were analyzed by a GLMM with treatment, visit, and treatment by visit interaction, and country as fixed effects. Comparison of response rates between each gefapixant treatment group and placebo was conducted using the stratified CMH test (stratified by country, unless stated otherwise). Missing data was categorized as discontinued or missing; Test type: Superiority or Other; p = 0.0031, Cochran-Mantel-Haenszel
Statistical Analysis 7: Comparison: Placebo vs Gefapixant 7.5 mg; Day 84: ≥30% Change: 7.5 mg gefapixant vs. placebo Cough frequency responder endpoints were analyzed by a GLMM with treatment, visit, and treatment by visit interaction, and country as fixed effects. Comparison of response rates between each gefapixant treatment group and placebo was conducted using the stratified CMH test (stratified by country, unless stated otherwise). Missing data was categorized as discontinued or missing; Test type: Superiority or Other; p = 0.0283, Cochran-Mantel-Haenszel
Statistical Analysis 8: Comparison: Placebo vs Gefapixant 20 mg; Day 84: ≥30% Change: 20 mg gefapixant vs. placebo Cough frequency responder endpoints were analyzed by a GLMM with treatment, visit, and treatment by visit interaction, and country as fixed effects. Comparison of response rates between each gefapixant treatment group and placebo was conducted using the stratified CMH test (stratified by country, unless stated otherwise). Missing data was categorized as discontinued or missing; Test type: Superiority or Other; p = 0.6233, Cochran-Mantel-Haenszel
Statistical Analysis 9: Comparison: Placebo vs Gefapixant 50 mg; Day 84: ≥30% Change: 50 mg gefapixant vs. placebo Cough frequency responder endpoints were analyzed by a GLMM with treatment, visit, and treatment by visit interaction, and country as fixed effects. Comparison of response rates between each gefapixant treatment group and placebo was conducted using the stratified CMH test (stratified by country, unless stated otherwise). Missing data was categorized as discontinued or missing; Test type: Superiority or Other; p = 0.0001, Cochran-Mantel-Haenszel

15. Secondary Outcome: Percentage of Participants With ≥70%, ≥50%, and ≥30% Change From Baseline in Awake Objective Cough Frequency at the Follow-up Visit (Day 98)
Description: Awake Objective Cough Frequency (per hour) was defined as the total number of cough events during the monitoring period (in general, 24-hr interval) while the participant was awake divided by the total duration (in hours) for the monitoring period that the participant was awake. 24 hour sound recordings were made at Baseline (Study Day -1) and at the Follow-up visit (Day 98) using a digital recording device. An independent cough monitoring center documented the time of each cough event over the 24 hour period, as well as the time when the participant went to sleep and the time the participant woke. The percentage of participants that met responder criteria for ≥70%, ≥50%, and ≥30% change (reduction) from baseline levels in Awake Objective Cough Frequency were reported for each treatment group at Day 98.
Time Frame: Baseline (Study Day -1), Day 98
Population: All randomized participants who had taken at least 1 dose of study medication and provided at least 1 baseline and at least one Day 98 endpoint observation during the treatment period.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Gefapixant 7.5 mg | Gefapixant 20 mg | Gefapixant 50 mg
Number analyzed (Participants) | 58 | 55 | 56 | 51
percentage of participants
  ≥70% Change | 13.8 (0.10) | 18.2 (0.10) | 14.3 (0.10) | 23.5 (0.10)
  ≥50% Change | 25.9 (0.11) | 32.7 (0.11) | 25.0 (0.11) | 39.2 (0.11)
  ≥30% Change | 51.7 (0.10) | 56.4 (0.10) | 50.0 (0.10) | 58.8 (0.11)
Statistical Analysis 1: Comparison: Placebo vs Gefapixant 7.5 mg; Day 98: ≥70% Change: 7.5 mg gefapixant vs. placebo Cough frequency responder endpoints were analyzed by a generalized linear mixed model (GLMM) with treatment, visit, and treatment by visit interaction, and country as fixed effects. Comparison of response rates between each gefapixant treatment group and placebo was conducted using the stratified Cochran Mantel Haenszel (CMH) test (stratified by country, unless stated otherwise). Missing data was categorized as discontinued or missing; Test type: Superiority or Other; p = 0.4925, Cochran-Mantel-Haenszel
Statistical Analysis 2: Comparison: Placebo vs Gefapixant 20 mg; Day 98: ≥70% Change: 20 mg gefapixant vs. placebo Cough frequency responder endpoints were analyzed by a GLMM with treatment, visit, and treatment by visit interaction, and country as fixed effects. Comparison of response rates between each gefapixant treatment group and placebo was conducted using the stratified CMH test (stratified by country, unless stated otherwise). Missing data was categorized as discontinued or missing; Test type: Superiority or Other; p = 0.9007, Cochran-Mantel-Haenszel
Statistical Analysis 3: Comparison: Placebo vs Gefapixant 50 mg; Day 98: ≥70% Change: 50 mg gefapixant vs. placebo Cough frequency responder endpoints were analyzed by a GLMM with treatment, visit, and treatment by visit interaction, and country as fixed effects. Comparison of response rates between each gefapixant treatment group and placebo was conducted using the stratified CMH test (stratified by country, unless stated otherwise). Missing data was categorized as discontinued or missing; Test type: Superiority or Other; p = 0.1602, Cochran-Mantel-Haenszel
Statistical Analysis 4: Comparison: Placebo vs Gefapixant 7.5 mg; Day 98: ≥50% Change: 7.5 mg gefapixant vs. placebo Cough frequency responder endpoints were analyzed by a GLMM with treatment, visit, and treatment by visit interaction, and country as fixed effects. Comparison of response rates between each gefapixant treatment group and placebo was conducted using the stratified CMH test (stratified by country, unless stated otherwise). Missing data was categorized as discontinued or missing; Test type: Superiority or Other; p = 0.3440, Cochran-Mantel-Haenszel
Statistical Analysis 5: Comparison: Placebo vs Gefapixant 20 mg; Day 98: ≥50% Change: 20 mg gefapixant vs. placebo Cough frequency responder endpoints were analyzed by a GLMM with treatment, visit, and treatment by visit interaction, and country as fixed effects. Comparison of response rates between each gefapixant treatment group and placebo was conducted using the stratified CMH test (stratified by country, unless stated otherwise). Missing data was categorized as discontinued or missing; Test type: Superiority or Other; p = 0.9876, Cochran-Mantel-Haenszel
Statistical Analysis 6: Comparison: Placebo vs Gefapixant 50 mg; Day 98: ≥50% Change: 50 mg gefapixant vs. placebo Cough frequency responder endpoints were analyzed by a GLMM with treatment, visit, and treatment by visit interaction, and country as fixed effects. Comparison of response rates between each gefapixant treatment group and placebo was conducted using the stratified CMH test (stratified by country, unless stated otherwise). Missing data was categorized as discontinued or missing; Test type: Superiority or Other; p = 0.0993, Cochran-Mantel-Haenszel
Statistical Analysis 7: Comparison: Placebo vs Gefapixant 7.5 mg; Day 98: ≥30% Change: 7.5 mg gefapixant vs. placebo Cough frequency responder endpoints were analyzed by a GLMM with treatment, visit, and treatment by visit interaction, and country as fixed effects. Comparison of response rates between each gefapixant treatment group and placebo was conducted using the stratified CMH test (stratified by country, unless stated otherwise). Missing data was categorized as discontinued or missing; Test type: Superiority or Other; p = 0.5968, Cochran-Mantel-Haenszel
Statistical Analysis 8: Comparison: Placebo vs Gefapixant 20 mg; Day 98: ≥30% Change: 20 mg gefapixant vs. placebo Cough frequency responder endpoints were analyzed by a GLMM with treatment, visit, and treatment by visit interaction, and country as fixed effects. Comparison of response rates between each gefapixant treatment group and placebo was conducted using the stratified CMH test (stratified by country, unless stated otherwise). Missing data was categorized as discontinued or missing; Test type: Superiority or Other; p = 0.8726, Cochran-Mantel-Haenszel
Statistical Analysis 9: Comparison: Placebo vs Gefapixant 50 mg; Day 98: ≥30% Change: 50 mg gefapixant vs. placebo Cough frequency responder endpoints were analyzed by a GLMM with treatment, visit, and treatment by visit interaction, and country as fixed effects. Comparison of response rates between each gefapixant treatment group and placebo was conducted using the stratified CMH test (stratified by country, unless stated otherwise). Missing data was categorized as discontinued or missing; Test type: Superiority or Other; p = 0.4092, Cochran-Mantel-Haenszel

16. Secondary Outcome: Percentage of Participants With ≥70%, ≥50%, and ≥30% Change From Baseline in 24-Hour Objective Cough Frequency After 4 Weeks of Treatment (Day 28)
Description: 24-hr Objective Cough Frequency was defined as the total number of cough events during the monitoring period divided by the total duration in hours for the monitoring period (generally 24 hours). 24 hour sound recordings were made at Baseline (Study Day -1) and at Week 4 (Day 28) using a digital recording device. An independent cough monitoring center documented the time of each cough event over the 24 hour period, as well as the time when the participant went to sleep and the time the participant woke. The percentage of participants that met responder criteria for ≥70%, ≥50%, and ≥30% change (reduction) from baseline levels in 24-hr Objective Cough Frequency were reported for each treatment group at Day 28.
Time Frame: Baseline (Study Day -1), Day 28
Population: as for outcome 12
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Gefapixant 7.5 mg | Gefapixant 20 mg | Gefapixant 50 mg
Number analyzed (Participants) | 60 | 55 | 59 | 55
percentage of participants
  ≥70% Change | 13.3 (0.10) | 25.5 (0.10) | 15.3 (0.10) | 34.5 (0.10)
  ≥50% Change | 21.7 (0.11) | 34.5 (0.11) | 30.5 (0.11) | 50.9 (0.11)
  ≥30% Change | 51.7 (0.10) | 58.2 (0.10) | 45.8 (0.10) | 67.3 (0.11)
Statistical Analysis 1: Comparison: Placebo vs Gefapixant 7.5 mg; [analysis description as in outcome 12, analysis 1]; Test type: Superiority or Other; p = 0.0781, Cochran-Mantel-Haenszel
Statistical Analysis 2: Comparison: Placebo vs Gefapixant 20 mg; [analysis description as in outcome 12, analysis 2]; Test type: Superiority or Other; p = 0.7098, Cochran-Mantel-Haenszel
Statistical Analysis 3: Comparison: Placebo vs Gefapixant 50 mg; [analysis description as in outcome 12, analysis 3]; Test type: Superiority or Other; p = 0.0068, Cochran-Mantel-Haenszel
Statistical Analysis 4: Comparison: Placebo vs Gefapixant 7.5 mg; [analysis description as in outcome 12, analysis 4]; Test type: Superiority or Other; p = 0.1284, Cochran-Mantel-Haenszel
Statistical Analysis 5: Comparison: Placebo vs Gefapixant 20 mg; [analysis description as in outcome 12, analysis 5]; Test type: Superiority or Other; p = 0.2670, Cochran-Mantel-Haenszel
Statistical Analysis 6: Comparison: Placebo vs Gefapixant 50 mg; [analysis description as in outcome 12, analysis 6]; Test type: Superiority or Other; p = 0.0013, Cochran-Mantel-Haenszel
Statistical Analysis 7: Comparison: Placebo vs Gefapixant 7.5 mg; [analysis description as in outcome 12, analysis 7]; Test type: Superiority or Other; p = 0.4343, Cochran-Mantel-Haenszel
Statistical Analysis 8: Comparison: Placebo vs Gefapixant 20 mg; [analysis description as in outcome 12, analysis 8]; Test type: Superiority or Other; p = 0.5384, Cochran-Mantel-Haenszel
Statistical Analysis 9: Comparison: Placebo vs Gefapixant 50 mg; [analysis description as in outcome 12, analysis 9]; Test type: Superiority or Other; p = 0.0822, Cochran-Mantel-Haenszel

17. Secondary Outcome: Percentage of Participants With ≥70%, ≥50%, and ≥30% Change From Baseline in 24-Hour Objective Cough Frequency After 8 Weeks of Treatment (Day 56)
Description: 24-hr Objective Cough Frequency was defined as the total number of cough events during the monitoring period divided by the total duration in hours for the monitoring period (generally 24 hours). 24 hour sound recordings were made at Baseline (Study Day -1) and at Week 8 (Day 56) using a digital recording device. An independent cough monitoring center documented the time of each cough event over the 24 hour period, as well as the time when the participant went to sleep and the time the participant woke. The percentage of participants that met responder criteria for ≥70%, ≥50%, and ≥30% change (reduction) from baseline levels in 24-hr Objective Cough Frequency were reported for each treatment group at Day 56.
Time Frame: Baseline (Study Day -1), Day 56
Population: as for outcome 13
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Gefapixant 7.5 mg | Gefapixant 20 mg | Gefapixant 50 mg
Number analyzed (Participants) | 57 | 56 | 59 | 51
percentage of participants
  ≥70% Change | 7.0 (0.10) | 32.1 (0.10) | 22.0 (0.10) | 37.3 (0.10)
  ≥50% Change | 28.1 (0.11) | 50.0 (0.11) | 32.2 (0.11) | 52.9 (0.11)
  ≥30% Change | 45.6 (0.10) | 62.5 (0.10) | 54.2 (0.10) | 78.4 (0.11)
Statistical Analysis 1: Comparison: Placebo vs Gefapixant 7.5 mg; [analysis description as in outcome 13, analysis 1]; Test type: Superiority or Other; p = 0.0006, Cochran-Mantel-Haenszel
Statistical Analysis 2: Comparison: Placebo vs Gefapixant 20 mg; [analysis description as in outcome 13, analysis 2]; Test type: Superiority or Other; p = 0.0223, Cochran-Mantel-Haenszel
Statistical Analysis 3: Comparison: Placebo vs Gefapixant 50 mg; [analysis description as in outcome 13, analysis 3]; Test type: Superiority or Other; p = 0.0001, Cochran-Mantel-Haenszel
Statistical Analysis 4: Comparison: Placebo vs Gefapixant 7.5 mg; [analysis description as in outcome 13, analysis 4]; Test type: Superiority or Other; p = 0.0165, Cochran-Mantel-Haenszel
Statistical Analysis 5: Comparison: Placebo vs Gefapixant 20 mg; [analysis description as in outcome 13, analysis 5]; Test type: Superiority or Other; p = 0.6255, Cochran-Mantel-Haenszel
Statistical Analysis 6: Comparison: Placebo vs Gefapixant 50 mg; [analysis description as in outcome 13, analysis 6]; Test type: Superiority or Other; p = 0.0085, Cochran-Mantel-Haenszel
Statistical Analysis 7: Comparison: Placebo vs Gefapixant 7.5 mg; [analysis description as in outcome 13, analysis 7]; Test type: Superiority or Other; p = 0.0722, Cochran-Mantel-Haenszel
Statistical Analysis 8: Comparison: Placebo vs Gefapixant 20 mg; [analysis description as in outcome 13, analysis 8]; Test type: Superiority or Other; p = 0.3577, Cochran-Mantel-Haenszel
Statistical Analysis 9: Comparison: Placebo vs Gefapixant 50 mg; [analysis description as in outcome 13, analysis 9]; Test type: Superiority or Other; p = 0.0006, Cochran-Mantel-Haenszel

18. Secondary Outcome: Percentage of Participants With ≥70%, ≥50%, and ≥30% Change From Baseline in 24-Hour Objective Cough Frequency After 12 Weeks of Treatment (Day 84)
Description: 24-hr Objective Cough Frequency was defined as the total number of cough events during the monitoring period divided by the total duration in hours for the monitoring period (generally 24 hours). 24 hour sound recordings were made at Baseline (Study Day -1) and at Week 12 (Day 84) using a digital recording device. An independent cough monitoring center documented the time of each cough event over the 24 hour period, as well as the time when the participant went to sleep and the time the participant woke. The percentage of participants that met responder criteria for ≥70%, ≥50%, and ≥30% change (reduction) from baseline levels in 24-hr Objective Cough Frequency were reported for each treatment group at Day 84.
Time Frame: Baseline (Study Day -1), Day 84
Population: as for outcome 14
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Gefapixant 7.5 mg | Gefapixant 20 mg | Gefapixant 50 mg
Number analyzed (Participants) | 57 | 56 | 56 | 51
percentage of participants
  ≥70% Change | 14.0 (0.10) | 19.6 (0.10) | 25.0 (0.10) | 31.4 (0.10)
  ≥50% Change | 24.6 (0.11) | 44.6 (0.11) | 32.1 (0.11) | 54.9 (0.11)
  ≥30% Change | 42.1 (0.10) | 62.5 (0.10) | 50.0 (0.10) | 78.4 (0.11)
Statistical Analysis 1: Comparison: Placebo vs Gefapixant 7.5 mg; [analysis description as in outcome 14, analysis 1]; Test type: Superiority or Other; p = 0.3845, Cochran-Mantel-Haenszel
Statistical Analysis 2: Comparison: Placebo vs Gefapixant 20 mg; [analysis description as in outcome 14, analysis 2]; Test type: Superiority or Other; p = 0.1177, Cochran-Mantel-Haenszel
Statistical Analysis 3: Comparison: Placebo vs Gefapixant 50 mg; [analysis description as in outcome 14, analysis 3]; Test type: Superiority or Other; p = 0.0236, Cochran-Mantel-Haenszel
Statistical Analysis 4: Comparison: Placebo vs Gefapixant 7.5 mg; [analysis description as in outcome 14, analysis 4]; Test type: Superiority or Other; p = 0.0192, Cochran-Mantel-Haenszel
Statistical Analysis 5: Comparison: Placebo vs Gefapixant 20 mg; [analysis description as in outcome 14, analysis 5]; Test type: Superiority or Other; p = 0.3301, Cochran-Mantel-Haenszel
Statistical Analysis 6: Comparison: Placebo vs Gefapixant 50 mg; [analysis description as in outcome 14, analysis 6]; Test type: Superiority or Other; p = 0.0008, Cochran-Mantel-Haenszel
Statistical Analysis 7: Comparison: Placebo vs Gefapixant 7.5 mg; [analysis description as in outcome 14, analysis 7]; Test type: Superiority or Other; p = 0.0285, Cochran-Mantel-Haenszel
Statistical Analysis 8: Comparison: Placebo vs Gefapixant 20 mg; [analysis description as in outcome 14, analysis 8]; Test type: Superiority or Other; p = 0.3856, Cochran-Mantel-Haenszel
Statistical Analysis 9: Comparison: Placebo vs Gefapixant 50 mg; [analysis description as in outcome 14, analysis 9]; Test type: Superiority or Other; p = 0.0001, Cochran-Mantel-Haenszel

19. Secondary Outcome: Percentage of Participants With ≥70%, ≥50%, and ≥30% Change From Baseline in 24-Hour Objective Cough Frequency at the Follow-up Visit (Day 98)
Description: 24-hr Objective Cough Frequency was defined as the total number of cough events during the monitoring period divided by the total duration in hours for the monitoring period (generally 24 hours). 24 hour sound recordings were made at Baseline (Study Day -1) and at Week 14 (Day 98) using a digital recording device. An independent cough monitoring center documented the time of each cough event over the 24 hour period, as well as the time when the participant went to sleep and the time the participant woke. The percentage of participants that met responder criteria for ≥70%, ≥50%, and ≥30% change (reduction) from baseline levels in 24-hr Objective Cough Frequency were reported for each treatment group at Day 98.
Time Frame: Baseline (Study Day -1), Day 98
Population: as for outcome 15
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Gefapixant 7.5 mg | Gefapixant 20 mg | Gefapixant 50 mg
Number analyzed (Participants) | 58 | 55 | 56 | 51
percentage of participants
  ≥70% Change | 12.1 (0.10) | 20.0 (0.10) | 16.1 (0.10) | 21.6 (0.10)
  ≥50% Change | 25.9 (0.11) | 34.5 (0.11) | 25.0 (0.11) | 39.2 (0.11)
  ≥30% Change | 46.6 (0.10) | 52.7 (0.10) | 46.4 (0.10) | 54.9 (0.11)
Statistical Analysis 1: Comparison: Placebo vs Gefapixant 7.5 mg; [analysis description as in outcome 15, analysis 1]; Test type: Superiority or Other; p = 0.2441, Cochran-Mantel-Haenszel
Statistical Analysis 2: Comparison: Placebo vs Gefapixant 20 mg; [analysis description as in outcome 15, analysis 2]; Test type: Superiority or Other; p = 0.5055, Cochran-Mantel-Haenszel
Statistical Analysis 3: Comparison: Placebo vs Gefapixant 50 mg; [analysis description as in outcome 15, analysis 3]; Test type: Superiority or Other; p = 0.1602, Cochran-Mantel-Haenszel
Statistical Analysis 4: Comparison: Placebo vs Gefapixant 7.5 mg; [analysis description as in outcome 15, analysis 4]; Test type: Superiority or Other; p = 0.2721, Cochran-Mantel-Haenszel
Statistical Analysis 5: Comparison: Placebo vs Gefapixant 20 mg; [analysis description as in outcome 15, analysis 5]; Test type: Superiority or Other; p = 0.9763, Cochran-Mantel-Haenszel
Statistical Analysis 6: Comparison: Placebo vs Gefapixant 50 mg; [analysis description as in outcome 15, analysis 6]; Test type: Superiority or Other; p = 0.0993, Cochran-Mantel-Haenszel
Statistical Analysis 7: Comparison: Placebo vs Gefapixant 7.5 mg; [analysis description as in outcome 15, analysis 7]; Test type: Superiority or Other; p = 0.4575, Cochran-Mantel-Haenszel
Statistical Analysis 8: Comparison: Placebo vs Gefapixant 20 mg; [analysis description as in outcome 15, analysis 8]; Test type: Superiority or Other; p = 0.9706, Cochran-Mantel-Haenszel
Statistical Analysis 9: Comparison: Placebo vs Gefapixant 50 mg; [analysis description as in outcome 15, analysis 9]; Test type: Superiority or Other; p = 0.3258, Cochran-Mantel-Haenszel

20. Secondary Outcome: Change From Baseline in Sleep Objective Cough Frequency After 4 Weeks of Treatment (Day 28)
Description: Sleep Objective Cough Frequency was defined as the total number of cough events during the monitoring period while the participant was asleep divided by the total duration in hours for the monitoring period that the participant was asleep. 24 hour sound recordings were made at Baseline (Study Day -1) and at Week 4 (Day 28) using a digital recording device. An independent cough monitoring center documented the time of each cough event over the 24 hour period, as well as the time when the participant went to sleep and the time the participant woke. LS mean change from baseline (in log scale) with associated SE reported for each treatment group. Change from Baseline in Sleep Objective Cough Frequency = (Post-Treatment Objective Sleep Cough Frequency minus Baseline Sleep Cough Frequency).
Time Frame: Baseline (Study Day -1), Day 28
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: log coughs/hour
Arm/Group | Placebo | Gefapixant 7.5 mg | Gefapixant 20 mg | Gefapixant 50 mg
Number analyzed (Participants) | 61 | 59 | 59 | 57
log coughs/hour | -0.37 (0.19) | -0.37 (0.20) | -0.38 (0.19) | -0.49 (0.20)
Statistical Analysis 1: Comparison: Placebo vs Gefapixant 7.5 mg; Day 28 Sleep Cough Frequency: 7.5 mg gefapixant vs. placebo Day 28 estimated treatment differences (gefapixant vs. placebo) and corresponding 95% CIs were estimated using a MMRM model, which included fixed effects for treatment group, visit, country, treatment-by-visit interaction, and Baseline value (on log scale) as a covariate; Test type: Other; p = 0.9858, Mixed Effect Repeated Measures model; LS Mean Difference = 0.00, 95% CI 2-sided [-0.53 to 0.54]
Statistical Analysis 2: Comparison: Placebo vs Gefapixant 20 mg; Day 28 Sleep Cough Frequency: 20 mg gefapixant vs. placebo Day 28 estimated treatment differences (gefapixant vs. placebo) and corresponding 95% CIs were estimated using a MMRM model, which included fixed effects for treatment group, visit, country, treatment-by-visit interaction, and Baseline value (on log scale) as a covariate; Test type: Other; p = 0.9813, Mixed Effect Repeated Measures model; LS Mean Difference = -0.01, 95% CI 2-sided [-0.53 to 0.52]
Statistical Analysis 3: Comparison: Placebo vs Gefapixant 50 mg; Day 28 Sleep Cough Frequency: 50 mg gefapixant vs. placebo Day 28 estimated treatment differences (gefapixant vs. placebo) and corresponding 95% CIs were estimated using a MMRM model, which included fixed effects for treatment group, visit, country, treatment-by-visit interaction, and Baseline value (on log scale) as a covariate; Test type: Other; p = 0.6746, Mixed Effect Repeated Measures model; LS Mean Difference = -0.11, 95% CI 2-sided [-0.65 to 0.42]

21. Secondary Outcome: Change From Baseline in Sleep Objective Cough Frequency After 8 Weeks of Treatment (Day 56)
Description: Sleep Objective Cough Frequency was defined as the total number of cough events during the monitoring period while the participant was asleep divided by the total duration in hours for the monitoring period that the participant was asleep. 24 hour sound recordings were made at Baseline (Study Day -1) and at Week 8 (Day 56) using a digital recording device. An independent cough monitoring center documented the time of each cough event over the 24 hour period, as well as the time when the participant went to sleep and the time the participant woke. LS mean change from baseline (in log scale) with associated SE reported for each treatment group. Change from Baseline in Sleep Objective Cough Frequency = (Post-Treatment Objective Sleep Cough Frequency minus Baseline Sleep Cough Frequency).
Time Frame: Baseline (Study Day -1), Day 56
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: log coughs/hour
Arm/Group | Placebo | Gefapixant 7.5 mg | Gefapixant 20 mg | Gefapixant 50 mg
Number analyzed (Participants) | 61 | 59 | 59 | 57
log coughs/hour | -0.40 (0.20) | -0.72 (0.20) | -0.40 (0.20) | -0.80 (0.21)
Statistical Analysis 1: Comparison: Placebo vs Gefapixant 7.5 mg; Day 56 Sleep Cough Frequency: 7.5 mg gefapixant vs. placebo Day 56 estimated treatment differences (gefapixant vs. placebo) and corresponding 95% CIs were estimated using a MMRM model, which included fixed effects for treatment group, visit, country, treatment-by-visit interaction, and Baseline value (on log scale) as a covariate; Test type: Other; p = 0.2583, Mixed Effect Repeated Measures model; LS Mean Difference = -0.32, 95% CI 2-sided [-0.88 to 0.24]
Statistical Analysis 2: Comparison: Placebo vs Gefapixant 20 mg; Day 56 Sleep Cough Frequency: 20 mg gefapixant vs. placebo Day 56 estimated treatment differences (gefapixant vs. placebo) and corresponding 95% CIs were estimated using a MMRM model, which included fixed effects for treatment group, visit, country, treatment-by-visit interaction, and Baseline value (on log scale) as a covariate; Test type: Other; p = 0.9826, Mixed Effect Repeated Measures model; LS Mean Difference = 0.01, 95% CI 2-sided [-0.55 to 0.56]
Statistical Analysis 3: Comparison: Placebo vs Gefapixant 50 mg; Day 56 Sleep Cough Frequency: 50 mg gefapixant vs. placebo Day 56 estimated treatment differences (gefapixant vs. placebo) and corresponding 95% CIs were estimated using a MMRM model, which included fixed effects for treatment group, visit, country, treatment-by-visit interaction, and Baseline value (on log scale) as a covariate; Test type: Other; p = 0.1672, Mixed Effect Repeated Measures model; LS Mean Difference = -0.40, 95% CI 2-sided [-0.98 to 0.17]

22. Secondary Outcome: Change From Baseline in Sleep Objective Cough Frequency After 12 Weeks of Treatment (Day 84)
Description: Sleep Objective Cough Frequency was defined as the total number of cough events during the monitoring period while the participant was asleep divided by the total duration in hours for the monitoring period that the participant was asleep. 24 hour sound recordings were made at Baseline (Study Day -1) and at Week 12 (Day 84) using a digital recording device. An independent cough monitoring center documented the time of each cough event over the 24 hour period, as well as the time when the participant went to sleep and the time the participant woke. LS mean change from baseline (in log scale) with associated SE reported for each treatment group. Change from Baseline in Sleep Objective Cough Frequency = (Post-Treatment Objective Sleep Cough Frequency minus Baseline Sleep Cough Frequency).
Time Frame: Baseline (Study Day -1), Day 84
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: log coughs/hour
Arm/Group | Placebo | Gefapixant 7.5 mg | Gefapixant 20 mg | Gefapixant 50 mg
Number analyzed (Participants) | 61 | 59 | 59 | 57
log coughs/hour | -0.72 (0.19) | -0.58 (0.20) | -0.65 (0.19) | -0.44 (0.20)
Statistical Analysis 1: Comparison: Placebo vs Gefapixant 7.5 mg; Day 84 Sleep Cough Frequency: 7.5 mg gefapixant vs. placebo Day 84 estimated treatment differences (gefapixant vs. placebo) and corresponding 95% CIs were estimated using a MMRM model, which included fixed effects for treatment group, visit, country, treatment-by-visit interaction, and Baseline value (on log scale) as a covariate; Test type: Other; p = 0.6102, Mixed Effect Repeated Measures model; LS Mean Difference = 0.14, 95% CI 2-sided [-0.4 to 0.68]
Statistical Analysis 2: Comparison: Placebo vs Gefapixant 20 mg; Day 84 Sleep Cough Frequency: 20 mg gefapixant vs. placebo Day 84 estimated treatment differences (gefapixant vs. placebo) and corresponding 95% CIs were estimated using a MMRM model, which included fixed effects for treatment group, visit, country, treatment-by-visit interaction, and Baseline value (on log scale) as a covariate; Test type: Other; p = 0.7782, Mixed Effect Repeated Measures model; LS Mean Difference = 0.08, 95% CI 2-sided [-0.46 to 0.61]
Statistical Analysis 3: Comparison: Placebo vs Gefapixant 50 mg; Day 84 Sleep Cough Frequency: 50 mg gefapixant vs. placebo Day 84 estimated treatment differences (gefapixant vs. placebo) and corresponding 95% CIs were estimated using a MMRM model, which included fixed effects for treatment group, visit, country, treatment-by-visit interaction, and Baseline value (on log scale) as a covariate; Test type: Other; p = 0.3167, Mixed Effect Repeated Measures model; LS Mean Difference = 0.28, 95% CI 2-sided [-0.27 to 0.83]

23. Secondary Outcome: Change From Baseline in Weekly Mean Daily Cough Severity Diary (CSD) Total Score at Week 1
Description: The daily CSD instrument has a total of 7 items, each with scores ranging from 0 (best) to 10 (worst). The total daily CSD is the sum of these 7 item scores (Min=0, Max=70). Mean total daily score (the sum of 7 item scores divided by 7) was derived for each day. Weekly mean total daily score was defined as the average of the mean total daily scores for each week. LS mean change from baseline of the weekly mean total daily CSD score was reported for each treatment group with associated SE. Baseline was defined as the average CSD scores collected during the week prior to Day 1 (Study Day -7 to Day -1).
Time Frame: Baseline, Week 1
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Gefapixant 7.5 mg | Gefapixant 20 mg | Gefapixant 50 mg
Number analyzed (Participants) | 61 | 59 | 59 | 57
score on a scale | -1.0 (0.15) | -0.7 (0.15) | -0.7 (0.15) | -1.0 (0.15)
Statistical Analysis 1: Comparison: Placebo vs Gefapixant 7.5 mg; Week 1 CSD Total Score: 7.5 mg gefapixant vs. placebo Week 1 estimated treatment differences (gefapixant vs. placebo) and corresponding 95% CIs were estimated using a MMRM model, which included fixed effects for treatment group, visit, country, treatment-by-visit interaction, and Baseline value as a covariate; Test type: Other; p = 0.1545, Mixed Effect Repeated Measures model; LS Mean Difference = 0.3, 95% CI 2-sided [-0.1 to 0.7]
Statistical Analysis 2: Comparison: Placebo vs Gefapixant 20 mg; Week 1 CSD Total Score: 20 mg gefapixant vs. placebo Week 1 estimated treatment differences (gefapixant vs. placebo) and corresponding 95% CIs were estimated using a MMRM model, which included fixed effects for treatment group, visit, country, treatment-by-visit interaction, and Baseline value as a covariate; Test type: Other; p = 0.2013, Mixed Effect Repeated Measures model; LS Mean Difference = 0.3, 95% CI 2-sided [-0.1 to 0.7]
Statistical Analysis 3: Comparison: Placebo vs Gefapixant 50 mg; Week 1 CSD Total Score: 50 mg gefapixant vs. placebo Week 1 estimated treatment differences (gefapixant vs. placebo) and corresponding 95% CIs were estimated using a MMRM model, which included fixed effects for treatment group, visit, country, treatment-by-visit interaction, and Baseline value as a covariate; Test type: Other; p = 0.9962, Mixed Effect Repeated Measures model; LS Mean Difference = 0.0, 95% CI 2-sided [-0.4 to 0.4]

24. Secondary Outcome: Change From Baseline in Weekly Mean Daily CSD Total Score at Week 2
Description: as for outcome 23
Time Frame: Baseline, Week 2
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Gefapixant 7.5 mg | Gefapixant 20 mg | Gefapixant 50 mg
Number analyzed (Participants) | 61 | 59 | 59 | 57
score on a scale | -1.0 (0.18) | -0.9 (0.19) | -1.0 (0.19) | -1.5 (0.19)
Statistical Analysis 1: Comparison: Placebo vs Gefapixant 7.5 mg; Week 2 CSD Total Score: 7.5 mg gefapixant vs. placebo Week 2 estimated treatment differences (gefapixant vs. placebo) and corresponding 95% CIs were estimated using a MMRM model, which included fixed effects for treatment group, visit, country, treatment-by-visit interaction, and Baseline value as a covariate; Test type: Other; p = 0.7328, Mixed Effect Repeated Measures model; LS Mean Difference = 0.1, 95% CI 2-sided [-0.4 to 0.6]
Statistical Analysis 2: Comparison: Placebo vs Gefapixant 20 mg; Week 2 CSD Total Score: 20 mg gefapixant vs. placebo Week 2 estimated treatment differences (gefapixant vs. placebo) and corresponding 95% CIs were estimated using a MMRM model, which included fixed effects for treatment group, visit, country, treatment-by-visit interaction, and Baseline value as a covariate; Test type: Other; p = 0.7635, Mixed Effect Repeated Measures model; LS Mean Difference = 0.1, 95% CI 2-sided [-0.4 to 0.6]
Statistical Analysis 3: Comparison: Placebo vs Gefapixant 50 mg; Week 2 CSD Total Score: 50 mg gefapixant vs. placebo Week 2 estimated treatment differences (gefapixant vs. placebo) and corresponding 95% CIs were estimated using a MMRM model, which included fixed effects for treatment group, visit, country, treatment-by-visit interaction, and Baseline value as a covariate; Test type: Other; p = 0.0951, Mixed Effect Repeated Measures model; LS Mean Difference = -0.4, 95% CI 2-sided [-0.9 to 0.1]

25. Secondary Outcome: Change From Baseline in Weekly Mean Daily CSD Total Score at Week 3
Description: as for outcome 23
Time Frame: Baseline, Week 3
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Gefapixant 7.5 mg | Gefapixant 20 mg | Gefapixant 50 mg
Number analyzed (Participants) | 61 | 59 | 59 | 57
score on a scale | -1.0 (0.20) | -1.2 (0.20) | -1.3 (0.20) | -1.5 (0.20)
Statistical Analysis 1: Comparison: Placebo vs Gefapixant 7.5 mg; Week 3 CSD Total Score: 7.5 mg gefapixant vs. placebo Week 3 estimated treatment differences (gefapixant vs. placebo) and corresponding 95% CIs were estimated using a MMRM model, which included fixed effects for treatment group, visit, country, treatment-by-visit interaction, and Baseline value as a covariate; Test type: Other; p = 0.5797, Mixed Effect Repeated Measures model; LS Mean Difference = -0.2, 95% CI 2-sided [-0.7 to 0.4]
Statistical Analysis 2: Comparison: Placebo vs Gefapixant 20 mg; Week 3 CSD Total Score: 20 mg gefapixant vs. placebo Week 3 estimated treatment differences (gefapixant vs. placebo) and corresponding 95% CIs were estimated using a MMRM model, which included fixed effects for treatment group, visit, country, treatment-by-visit interaction, and Baseline value as a covariate; Test type: Other; p = 0.2499, Mixed Effect Repeated Measures model; LS Mean Difference = -0.3, 95% CI 2-sided [-0.9 to 0.2]
Statistical Analysis 3: Comparison: Placebo vs Gefapixant 50 mg; Week 3 CSD Total Score: 50 mg gefapixant vs. placebo Week 3 estimated treatment differences (gefapixant vs. placebo) and corresponding 95% CIs were estimated using a MMRM model, which included fixed effects for treatment group, visit, country, treatment-by-visit interaction, and Baseline value as a covariate; Test type: Other; p = 0.0612, Mixed Effect Repeated Measures model; LS Mean Difference = -0.5, 95% CI 2-sided [-1.1 to 0.0]

26. Secondary Outcome: Change From Baseline in Weekly Mean Daily CSD Total Score at Week 4
Description: as for outcome 23
Time Frame: Baseline, Week 4
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Gefapixant 7.5 mg | Gefapixant 20 mg | Gefapixant 50 mg
Number analyzed (Participants) | 61 | 59 | 59 | 57
score on a scale | -1.2 (0.20) | -1.4 (0.20) | -1.5 (0.20) | -1.7 (0.20)
Statistical Analysis 1: Comparison: Placebo vs Gefapixant 7.5 mg; Week 4 CSD Total Score: 7.5 mg gefapixant vs. placebo Week 4 estimated treatment differences (gefapixant vs. placebo) and corresponding 95% CIs were estimated using a MMRM model, which included fixed effects for treatment group, visit, country, treatment-by-visit interaction, and Baseline value as a covariate; Test type: Other; p = 0.5358, Mixed Effect Repeated Measures model; LS Mean Difference = -0.2, 95% CI 2-sided [-0.7 to 0.4]
Statistical Analysis 2: Comparison: Placebo vs Gefapixant 20 mg; Week 4 CSD Total Score: 20 mg gefapixant vs. placebo Week 4 estimated treatment differences (gefapixant vs. placebo) and corresponding 95% CIs were estimated using a MMRM model, which included fixed effects for treatment group, visit, country, treatment-by-visit interaction, and Baseline value as a covariate; Test type: Other; p = 0.3129, Mixed Effect Repeated Measures model; LS Mean Difference = -0.3, 95% CI 2-sided [-0.8 to 0.3]
Statistical Analysis 3: Comparison: Placebo vs Gefapixant 50 mg; Week 4 CSD Total Score: 50 mg gefapixant vs. placebo Week 4 estimated treatment differences (gefapixant vs. placebo) and corresponding 95% CIs were estimated using a MMRM model, which included fixed effects for treatment group, visit, country, treatment-by-visit interaction, and Baseline value as a covariate; Test type: Other; p = 0.1046, Mixed Effect Repeated Measures model; LS Mean Difference = -0.5, 95% CI 2-sided [-1.0 to 0.1]

27. Secondary Outcome: Change From Baseline in Weekly Mean Daily CSD Total Score at Week 5
Description: as for outcome 23
Time Frame: Baseline, Week 5
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Gefapixant 7.5 mg | Gefapixant 20 mg | Gefapixant 50 mg
Number analyzed (Participants) | 61 | 59 | 59 | 57
score on a scale | -1.1 (0.20) | -1.3 (0.20) | -1.5 (0.20) | -1.8 (0.21)
Statistical Analysis 1: Comparison: Placebo vs Gefapixant 7.5 mg; Week 5 CSD Total Score: 7.5 mg gefapixant vs. placebo Week 5 estimated treatment differences (gefapixant vs. placebo) and corresponding 95% CIs were estimated using a MMRM model, which included fixed effects for treatment group, visit, country, treatment-by-visit interaction, and Baseline value as a covariate; Test type: Other; p = 0.5796, Mixed Effect Repeated Measures model; LS Mean Difference = -0.2, 95% CI 2-sided [-0.7 to 0.4]
Statistical Analysis 2: Comparison: Placebo vs Gefapixant 20 mg; Week 5 CSD Total Score: 20 mg gefapixant vs. placebo Week 5 estimated treatment differences (gefapixant vs. placebo) and corresponding 95% CIs were estimated using a MMRM model, which included fixed effects for treatment group, visit, country, treatment-by-visit interaction, and Baseline value as a covariate; Test type: Other; p = 0.1430, Mixed Effect Repeated Measures model; LS Mean Difference = -0.4, 95% CI 2-sided [-1.0 to 0.1]
Statistical Analysis 3: Comparison: Placebo vs Gefapixant 50 mg; Week 5 CSD Total Score: 50 mg gefapixant vs. placebo Week 5 estimated treatment differences (gefapixant vs. placebo) and corresponding 95% CIs were estimated using a MMRM model, which included fixed effects for treatment group, visit, country, treatment-by-visit interaction, and Baseline value as a covariate; Test type: Other; p = 0.0221, Mixed Effect Repeated Measures model; LS Mean Difference = -0.7, 95% CI 2-sided [-1.2 to -0.1]

28. Secondary Outcome: Change From Baseline in Weekly Mean Daily CSD Total Score at Week 6
Description: as for outcome 23
Time Frame: Baseline, Week 6
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Gefapixant 7.5 mg | Gefapixant 20 mg | Gefapixant 50 mg
Number analyzed (Participants) | 61 | 59 | 59 | 57
score on a scale | -1.0 (0.21) | -1.4 (0.21) | -1.5 (0.21) | -1.7 (0.21)
Statistical Analysis 1: Comparison: Placebo vs Gefapixant 7.5 mg; Week 6 CSD Total Score: 7.5 mg gefapixant vs. placebo Week 6 estimated treatment differences (gefapixant vs. placebo) and corresponding 95% CIs were estimated using a MMRM model, which included fixed effects for treatment group, visit, country, treatment-by-visit interaction, and Baseline value as a covariate; Test type: Other; p = 0.1562, Mixed Effect Repeated Measures model; LS Mean Difference = -0.4, 95% CI 2-sided [-1.0 to 0.2]
Statistical Analysis 2: Comparison: Placebo vs Gefapixant 20 mg; Week 6 CSD Total Score: 20 mg gefapixant vs. placebo Week 6 estimated treatment differences (gefapixant vs. placebo) and corresponding 95% CIs were estimated using a MMRM model, which included fixed effects for treatment group, visit, country, treatment-by-visit interaction, and Baseline value as a covariate; Test type: Other; p = 0.0710, Mixed Effect Repeated Measures model; LS Mean Difference = -0.5, 95% CI 2-sided [-1.1 to 0.0]
Statistical Analysis 3: Comparison: Placebo vs Gefapixant 50 mg; Week 6 CSD Total Score: 50 mg gefapixant vs. placebo Week 6 estimated treatment differences (gefapixant vs. placebo) and corresponding 95% CIs were estimated using a MMRM model, which included fixed effects for treatment group, visit, country, treatment-by-visit interaction, and Baseline value as a covariate; Test type: Other; p = 0.0274, Mixed Effect Repeated Measures model; LS Mean Difference = -0.7, 95% CI 2-sided [-1.2 to -0.1]

29. Secondary Outcome: Change From Baseline in Weekly Mean Daily CSD Total Score at Week 7
Description: as for outcome 23
Time Frame: Baseline, Week 7
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Gefapixant 7.5 mg | Gefapixant 20 mg | Gefapixant 50 mg
Number analyzed (Participants) | 61 | 59 | 59 | 57
score on a scale | -1.2 (0.21) | -1.4 (0.22) | -1.5 (0.22) | -1.7 (0.22)
Statistical Analysis 1: Comparison: Placebo vs Gefapixant 7.5 mg; Week 7 CSD Total Score: 7.5 mg gefapixant vs. placebo Week 7 estimated treatment differences (gefapixant vs. placebo) and corresponding 95% CIs were estimated using a MMRM model, which included fixed effects for treatment group, visit, country, treatment-by-visit interaction, and Baseline value as a covariate; Test type: Other; p = 0.4464, Mixed Effect Repeated Measures model; LS Mean Difference = -0.2, 95% CI 2-sided [-0.8 to 0.4]
Statistical Analysis 2: Comparison: Placebo vs Gefapixant 20 mg; Week 7 CSD Total Score: 20 mg gefapixant vs. placebo Week 7 estimated treatment differences (gefapixant vs. placebo) and corresponding 95% CIs were estimated using a MMRM model, which included fixed effects for treatment group, visit, country, treatment-by-visit interaction, and Baseline value as a covariate; Test type: Other; p = 0.3320, Mixed Effect Repeated Measures model; LS Mean Difference = -0.3, 95% CI 2-sided [-0.9 to 0.3]
Statistical Analysis 3: Comparison: Placebo vs Gefapixant 50 mg; Week 7 CSD Total Score: 50 mg gefapixant vs. placebo Week 7 estimated treatment differences (gefapixant vs. placebo) and corresponding 95% CIs were estimated using a MMRM model, which included fixed effects for treatment group, visit, country, treatment-by-visit interaction, and Baseline value as a covariate; Test type: Other; p = 0.0792, Mixed Effect Repeated Measures model; LS Mean Difference = -0.5, 95% CI 2-sided [-1.1 to 0.1]

30. Secondary Outcome: Change From Baseline in Weekly Mean Daily CSD Total Score at Week 8
Description: as for outcome 23
Time Frame: Baseline, Week 8
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Gefapixant 7.5 mg | Gefapixant 20 mg | Gefapixant 50 mg
Number analyzed (Participants) | 61 | 59 | 59 | 57
score on a scale | -1.3 (0.22) | -1.5 (0.22) | -1.6 (0.22) | -1.7 (0.23)
Statistical Analysis 1: Comparison: Placebo vs Gefapixant 7.5 mg; Week 8 CSD Total Score: 7.5 mg gefapixant vs. placebo Week 8 estimated treatment differences (gefapixant vs. placebo) and corresponding 95% CIs were estimated using a MMRM model, which included fixed effects for treatment group, visit, country, treatment-by-visit interaction, and Baseline value as a covariate; Test type: Other; p = 0.4716, Mixed Effect Repeated Measures model; LS Mean Difference = -0.2, 95% CI 2-sided [-0.8 to 0.4]
Statistical Analysis 2: Comparison: Placebo vs Gefapixant 20 mg; Week 8 CSD Total Score: 20 mg gefapixant vs. placebo Week 8 estimated treatment differences (gefapixant vs. placebo) and corresponding 95% CIs were estimated using a MMRM model, which included fixed effects for treatment group, visit, country, treatment-by-visit interaction, and Baseline value as a covariate; Test type: Other; p = 0.4371, Mixed Effect Repeated Measures model; LS Mean Difference = -0.2, 95% CI 2-sided [-0.8 to 0.4]
Statistical Analysis 3: Comparison: Placebo vs Gefapixant 50 mg; Week 8 CSD Total Score: 50 mg gefapixant vs. placebo Week 8 estimated treatment differences (gefapixant vs. placebo) and corresponding 95% CIs were estimated using a MMRM model, which included fixed effects for treatment group, visit, country, treatment-by-visit interaction, and Baseline value as a covariate; Test type: Other; p = 0.1907, Mixed Effect Repeated Measures model; LS Mean Difference = -0.4, 95% CI 2-sided [-1.0 to 0.2]

31. Secondary Outcome: Change From Baseline in Weekly Mean Daily CSD Total Score at Week 9
Description: as for outcome 23
Time Frame: Baseline, Week 9
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Gefapixant 7.5 mg | Gefapixant 20 mg | Gefapixant 50 mg
Number analyzed (Participants) | 61 | 59 | 59 | 57
score on a scale | -1.3 (0.21) | -1.6 (0.22) | -1.7 (0.22) | -1.8 (0.22)
Statistical Analysis 1: Comparison: Placebo vs Gefapixant 7.5 mg; Week 9 CSD Total Score: 7.5 mg gefapixant vs. placebo Week 9 estimated treatment differences (gefapixant vs. placebo) and corresponding 95% CIs were estimated using a MMRM model, which included fixed effects for treatment group, visit, country, treatment-by-visit interaction, and Baseline value as a covariate; Test type: Other; p = 0.2772, Mixed Effect Repeated Measures model; LS Mean Difference = -0.3, 95% CI 2-sided [-0.9 to 0.3]
Statistical Analysis 2: Comparison: Placebo vs Gefapixant 20 mg; Week 9 CSD Total Score: 20 mg gefapixant vs. placebo Week 9 estimated treatment differences (gefapixant vs. placebo) and corresponding 95% CIs were estimated using a MMRM model, which included fixed effects for treatment group, visit, country, treatment-by-visit interaction, and Baseline value as a covariate; Test type: Other; p = 0.1132, Mixed Effect Repeated Measures model; LS Mean Difference = -0.5, 95% CI 2-sided [-1.1 to 0.1]
Statistical Analysis 3: Comparison: Placebo vs Gefapixant 50 mg; Week 9 CSD Total Score: 50 mg gefapixant vs. placebo Week 9 estimated treatment differences (gefapixant vs. placebo) and corresponding 95% CIs were estimated using a MMRM model, which included fixed effects for treatment group, visit, country, treatment-by-visit interaction, and Baseline value as a covariate; Test type: Other; p = 0.0737, Mixed Effect Repeated Measures model; LS Mean Difference = -0.6, 95% CI 2-sided [-1.2 to 0.1]

32. Secondary Outcome: Change From Baseline in Weekly Mean Daily CSD Total Score at Week 10
Description: as for outcome 23
Time Frame: Baseline, Week 10
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Gefapixant 7.5 mg | Gefapixant 20 mg | Gefapixant 50 mg
Number analyzed (Participants) | 61 | 59 | 59 | 57
score on a scale | -1.2 (0.22) | -1.4 (0.22) | -1.6 (0.22) | -1.9 (0.22)
Statistical Analysis 1: Comparison: Placebo vs Gefapixant 7.5 mg; Week 10 CSD Total Score: 7.5 mg gefapixant vs. placebo Week 10 estimated treatment differences (gefapixant vs. placebo) and corresponding 95% CIs were estimated using a MMRM model, which included fixed effects for treatment group, visit, country, treatment-by-visit interaction, and Baseline value as a covariate; Test type: Other; p = 0.6266, Mixed Effect Repeated Measures model; LS Mean Difference = -0.1, 95% CI 2-sided [-0.8 to 0.5]
Statistical Analysis 2: Comparison: Placebo vs Gefapixant 20 mg; Week 10 CSD Total Score: 20 mg gefapixant vs. placebo Week 10 estimated treatment differences (gefapixant vs. placebo) and corresponding 95% CIs were estimated using a MMRM model, which included fixed effects for treatment group, visit, country, treatment-by-visit interaction, and Baseline value as a covariate; Test type: Other; p = 0.1769, Mixed Effect Repeated Measures model; LS Mean Difference = -0.4, 95% CI 2-sided [-1.0 to 0.2]
Statistical Analysis 3: Comparison: Placebo vs Gefapixant 50 mg; Week 10 CSD Total Score: 50 mg gefapixant vs. placebo Week 10 estimated treatment differences (gefapixant vs. placebo) and corresponding 95% CIs were estimated using a MMRM model, which included fixed effects for treatment group, visit, country, treatment-by-visit interaction, and Baseline value as a covariate; Test type: Other; p = 0.0313, Mixed Effect Repeated Measures model; LS Mean Difference = -0.7, 95% CI 2-sided [-1.3 to -0.1]

33. Secondary Outcome: Change From Baseline in Weekly Mean Daily CSD Total Score at Week 11
Description: as for outcome 23
Time Frame: Baseline, Week 11
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Gefapixant 7.5 mg | Gefapixant 20 mg | Gefapixant 50 mg
Number analyzed (Participants) | 61 | 59 | 59 | 57
score on a scale | -1.1 (0.22) | -1.5 (0.22) | -1.7 (0.22) | -1.9 (0.23)
Statistical Analysis 1: Comparison: Placebo vs Gefapixant 7.5 mg; Week 11 CSD Total Score: 7.5 mg gefapixant vs. placebo Week 11 estimated treatment differences (gefapixant vs. placebo) and corresponding 95% CIs were estimated using a MMRM model, which included fixed effects for treatment group, visit, country, treatment-by-visit interaction, and Baseline value as a covariate; Test type: Other; p = 0.2058, Mixed Effect Repeated Measures model; LS Mean Difference = -0.4, 95% CI 2-sided [-1.0 to 0.2]
Statistical Analysis 2: Comparison: Placebo vs Gefapixant 20 mg; Week 11 CSD Total Score: 20 mg gefapixant vs. placebo Week 11 estimated treatment differences (gefapixant vs. placebo) and corresponding 95% CIs were estimated using a MMRM model, which included fixed effects for treatment group, visit, country, treatment-by-visit interaction, and Baseline value as a covariate; Test type: Other; p = 0.0665, Mixed Effect Repeated Measures model; LS Mean Difference = -0.6, 95% CI 2-sided [-1.2 to 0.0]
Statistical Analysis 3: Comparison: Placebo vs Gefapixant 50 mg; Week 11 CSD Total Score: 50 mg gefapixant vs. placebo Week 11 estimated treatment differences (gefapixant vs. placebo) and corresponding 95% CIs were estimated using a MMRM model, which included fixed effects for treatment group, visit, country, treatment-by-visit interaction, and Baseline value as a covariate; Test type: Other; p = 0.0155, Mixed Effect Repeated Measures model; LS Mean Difference = -0.8, 95% CI 2-sided [-1.4 to -0.1]

34. Secondary Outcome: Change From Baseline in Weekly Mean Daily CSD Total Score at Week 12
Description: as for outcome 23
Time Frame: Baseline, Week 12
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Gefapixant 7.5 mg | Gefapixant 20 mg | Gefapixant 50 mg
Number analyzed (Participants) | 61 | 59 | 59 | 57
score on a scale | -1.2 (0.22) | -1.5 (0.22) | -1.7 (0.22) | -1.9 (0.23)
Statistical Analysis 1: Comparison: Placebo vs Gefapixant 7.5 mg; Week 12 CSD Total Score: 7.5 mg gefapixant vs. placebo Week 12 estimated treatment differences (gefapixant vs. placebo) and corresponding 95% CIs were estimated using a MMRM model, which included fixed effects for treatment group, visit, country, treatment-by-visit interaction, and Baseline value as a covariate; Test type: Other; p = 0.2458, Mixed Effect Repeated Measures model; LS Mean Difference = -0.4, 95% CI 2-sided [-1.0 to 0.3]
Statistical Analysis 2: Comparison: Placebo vs Gefapixant 20 mg; Week 12 CSD Total Score: 20 mg gefapixant vs. placebo Week 12 estimated treatment differences (gefapixant vs. placebo) and corresponding 95% CIs were estimated using a MMRM model, which included fixed effects for treatment group, visit, country, treatment-by-visit interaction, and Baseline value as a covariate; Test type: Other; p = 0.0662, Mixed Effect Repeated Measures model; LS Mean Difference = -0.6, 95% CI 2-sided [-1.2 to 0.0]
Statistical Analysis 3: Comparison: Placebo vs Gefapixant 50 mg; Week 12 CSD Total Score: 50 mg gefapixant vs. placebo Week 12 estimated treatment differences (gefapixant vs. placebo) and corresponding 95% CIs were estimated using a MMRM model, which included fixed effects for treatment group, visit, country, treatment-by-visit interaction, and Baseline value as a covariate; Test type: Other; p = 0.0197, Mixed Effect Repeated Measures model; LS Mean Difference = -0.7, 95% CI 2-sided [-1.4 to -0.1]

35. Secondary Outcome: Change From Baseline in Weekly Mean Daily Cough Score (DCS) at Week 1
Description: The DCS has a score ranging from 0 (best) to 10 (worst). Weekly mean daily score was defined as the average of the daily scores for each week. Baseline was defined as the average DCS score collected during the week prior to Day 1 (Day -7 to Day -1). Participants rated the severity of their cough using the DCS each day. LS mean change from baseline of the weekly mean Daily Cough Score with associated SE was reported for each treatment group.
Time Frame: Baseline, Week 1
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Gefapixant 7.5 mg | Gefapixant 20 mg | Gefapixant 50 mg
Number analyzed (Participants) | 61 | 59 | 59 | 57
score on a scale | -1.1 (0.18) | -0.7 (0.18) | -0.8 (0.19) | -1.1 (0.19)
Statistical Analysis 1: Comparison: Placebo vs Gefapixant 7.5 mg; Week 1 DCS Total Score: 7.5 mg gefapixant vs. placebo Week 1 estimated treatment differences (gefapixant vs. placebo) and corresponding 95% CIs were estimated using a MMRM model, which included fixed effects for treatment group, visit, country, treatment-by-visit interaction, and Baseline value as a covariate; Test type: Other; p = 0.1921, Mixed Effect Repeated Measures model; LS Mean Difference = 0.3, 95% CI 2-sided [-0.2 to 0.8]
Statistical Analysis 2: Comparison: Placebo vs Gefapixant 20 mg; Week 1 DCS Total Score: 20 mg gefapixant vs. placebo Week 1 estimated treatment differences (gefapixant vs. placebo) and corresponding 95% CIs were estimated using a MMRM model, which included fixed effects for treatment group, visit, country, treatment-by-visit interaction, and Baseline value as a covariate; Test type: Other; p = 0.2428, Mixed Effect Repeated Measures model; LS Mean Difference = 0.3, 95% CI 2-sided [-0.2 to 0.8]
Statistical Analysis 3: Comparison: Placebo vs Gefapixant 50 mg; Week 1 DCS Total Score: 50 mg gefapixant vs. placebo Week 1 estimated treatment differences (gefapixant vs. placebo) and corresponding 95% CIs were estimated using a MMRM model, which included fixed effects for treatment group, visit, country, treatment-by-visit interaction, and Baseline value as a covariate; Test type: Other; p = 0.7383, Mixed Effect Repeated Measures model; LS Mean Difference = -0.1, 95% CI 2-sided [-0.6 to 0.4]

36. Secondary Outcome: Change From Baseline in Weekly Mean DCS at Week 2
Description: as for outcome 35
Time Frame: Baseline, Week 2
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Gefapixant 7.5 mg | Gefapixant 20 mg | Gefapixant 50 mg
Number analyzed (Participants) | 61 | 59 | 59 | 57
score on a scale | -1.4 (0.22) | -1.1 (0.23) | -1.1 (0.23) | -1.7 (0.23)
Statistical Analysis 1: Comparison: Placebo vs Gefapixant 7.5 mg; Week 2 DCS Total Score: 7.5 mg gefapixant vs. placebo Week 2 estimated treatment differences (gefapixant vs. placebo) and corresponding 95% CIs were estimated using a MMRM model, which included fixed effects for treatment group, visit, country, treatment-by-visit interaction, and Baseline value as a covariate; Test type: Other; p = 0.4033, Mixed Effect Repeated Measures model; LS Mean Difference = 0.3, 95% CI 2-sided [-0.4 to 0.9]
Statistical Analysis 2: Comparison: Placebo vs Gefapixant 20 mg; Week 2 DCS Total Score: 20 mg gefapixant vs. placebo Week 2 estimated treatment differences (gefapixant vs. placebo) and corresponding 95% CIs were estimated using a MMRM model, which included fixed effects for treatment group, visit, country, treatment-by-visit interaction, and Baseline value as a covariate; Test type: Other; p = 0.4599, Mixed Effect Repeated Measures model; LS Mean Difference = 0.2, 95% CI 2-sided [-0.4 to 0.9]
Statistical Analysis 3: Comparison: Placebo vs Gefapixant 50 mg; Week 2 DCS Total Score: 50 mg gefapixant vs. placebo Week 2 estimated treatment differences (gefapixant vs. placebo) and corresponding 95% CIs were estimated using a MMRM model, which included fixed effects for treatment group, visit, country, treatment-by-visit interaction, and Baseline value as a covariate; Test type: Other; p = 0.2837, Mixed Effect Repeated Measures model; LS Mean Difference = -0.3, 95% CI 2-sided [-1.0 to 0.3]

37. Secondary Outcome: Change From Baseline in Weekly Mean DCS at Week 3
Description: as for outcome 35
Time Frame: Baseline, Week 3
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Gefapixant 7.5 mg | Gefapixant 20 mg | Gefapixant 50 mg
Number analyzed (Participants) | 61 | 59 | 59 | 57
score on a scale | -1.4 (0.24) | -1.3 (0.24) | -1.6 (0.25) | -1.7 (0.25)
Statistical Analysis 1: Comparison: Placebo vs Gefapixant 7.5 mg; Week 3 DCS Total Score: 7.5 mg gefapixant vs. placebo Week 3 estimated treatment differences (gefapixant vs. placebo) and corresponding 95% CIs were estimated using a MMRM model, which included fixed effects for treatment group, visit, country, treatment-by-visit interaction, and Baseline value as a covariate; Test type: Other; p = 0.8084, Mixed Effect Repeated Measures model; LS Mean Difference = 0.1, 95% CI 2-sided [-0.6 to 0.8]
Statistical Analysis 2: Comparison: Placebo vs Gefapixant 20 mg; Week 3 DCS Total Score: 20 mg gefapixant vs. placebo Week 3 estimated treatment differences (gefapixant vs. placebo) and corresponding 95% CIs were estimated using a MMRM model, which included fixed effects for treatment group, visit, country, treatment-by-visit interaction, and Baseline value as a covariate; Test type: Other; p = 0.6108, Mixed Effect Repeated Measures model; LS Mean Difference = -0.2, 95% CI 2-sided [-0.8 to 0.5]
Statistical Analysis 3: Comparison: Placebo vs Gefapixant 50 mg; Week 3 DCS Total Score: 50 mg gefapixant vs. placebo Week 3 estimated treatment differences (gefapixant vs. placebo) and corresponding 95% CIs were estimated using a MMRM model, which included fixed effects for treatment group, visit, country, treatment-by-visit interaction, and Baseline value as a covariate; Test type: Other; p = 0.4220, Mixed Effect Repeated Measures model; LS Mean Difference = -0.3, 95% CI 2-sided [-0.9 to 0.4]

38. Secondary Outcome: Change From Baseline in Weekly Mean DCS at Week 4
Description: as for outcome 35
Time Frame: Baseline, Week 4
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Gefapixant 7.5 mg | Gefapixant 20 mg | Gefapixant 50 mg
Number analyzed (Participants) | 61 | 59 | 59 | 57
score on a scale | -1.5 (0.24) | -1.6 (0.24) | -1.8 (0.24) | -1.9 (0.24)
Statistical Analysis 1: Comparison: Placebo vs Gefapixant 7.5 mg; Week 4 DCS Total Score: 7.5 mg gefapixant vs. placebo Week 4 estimated treatment differences (gefapixant vs. placebo) and corresponding 95% CIs were estimated using a MMRM model, which included fixed effects for treatment group, visit, country, treatment-by-visit interaction, and Baseline value as a covariate; Test type: Other; p = 0.8457, Mixed Effect Repeated Measures model; LS Mean Difference = -0.1, 95% CI 2-sided [-0.7 to 0.6]
Statistical Analysis 2: Comparison: Placebo vs Gefapixant 20 mg; Week 4 DCS Total Score: 20 mg gefapixant vs. placebo Week 4 estimated treatment differences (gefapixant vs. placebo) and corresponding 95% CIs were estimated using a MMRM model, which included fixed effects for treatment group, visit, country, treatment-by-visit interaction, and Baseline value as a covariate; Test type: Other; p = 0.4044, Mixed Effect Repeated Measures model; LS Mean Difference = -0.3, 95% CI 2-sided [-0.9 to 0.4]
Statistical Analysis 3: Comparison: Placebo vs Gefapixant 50 mg; Week 4 DCS Total Score: 50 mg gefapixant vs. placebo Week 4 estimated treatment differences (gefapixant vs. placebo) and corresponding 95% CIs were estimated using a MMRM model, which included fixed effects for treatment group, visit, country, treatment-by-visit interaction, and Baseline value as a covariate; Test type: Other; p = 0.3031, Mixed Effect Repeated Measures model; LS Mean Difference = -0.3, 95% CI 2-sided [-1.0 to 0.3]

39. Secondary Outcome: Change From Baseline in Weekly Mean DCS at Week 5
Description: as for outcome 35
Time Frame: Baseline, Week 5
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Gefapixant 7.5 mg | Gefapixant 20 mg | Gefapixant 50 mg
Number analyzed (Participants) | 61 | 59 | 59 | 57
score on a scale | -1.4 (0.23) | -1.4 (0.24) | -1.9 (0.24) | -2.1 (0.24)
Statistical Analysis 1: Comparison: Placebo vs Gefapixant 7.5 mg; Week 5 DCS Total Score: 7.5 mg gefapixant vs. placebo Week 5 estimated treatment differences (gefapixant vs. placebo) and corresponding 95% CIs were estimated using a MMRM model, which included fixed effects for treatment group, visit, country, treatment-by-visit interaction, and Baseline value as a covariate; Test type: Other; p = 0.9126, Mixed Effect Repeated Measures model; LS Mean Difference = -0.0, 95% CI 2-sided [-0.7 to 0.6]
Statistical Analysis 2: Comparison: Placebo vs Gefapixant 20 mg; Week 5 DCS Total Score: 20 mg gefapixant vs. placebo Week 5 estimated treatment differences (gefapixant vs. placebo) and corresponding 95% CIs were estimated using a MMRM model, which included fixed effects for treatment group, visit, country, treatment-by-visit interaction, and Baseline value as a covariate; Test type: Other; p = 0.1136, Mixed Effect Repeated Measures model; LS Mean Difference = -0.5, 95% CI 2-sided [-1.2 to 0.1]
Statistical Analysis 3: Comparison: Placebo vs Gefapixant 50 mg; Week 5 DCS Total Score: 50 mg gefapixant vs. placebo Week 5 estimated treatment differences (gefapixant vs. placebo) and corresponding 95% CIs were estimated using a MMRM model, which included fixed effects for treatment group, visit, country, treatment-by-visit interaction, and Baseline value as a covariate; Test type: Other; p = 0.0352, Mixed Effect Repeated Measures model; LS Mean Difference = -0.7, 95% CI 2-sided [-1.4 to -0.0]

40. Secondary Outcome: Change From Baseline in Weekly Mean DCS at Week 6
Description: as for outcome 35
Time Frame: Baseline, Week 6
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Gefapixant 7.5 mg | Gefapixant 20 mg | Gefapixant 50 mg
Number analyzed (Participants) | 61 | 59 | 59 | 57
score on a scale | -1.2 (0.24) | -1.7 (0.24) | -1.9 (0.24) | -1.8 (0.24)
Statistical Analysis 1: Comparison: Placebo vs Gefapixant 7.5 mg; Week 6 DCS Total Score: 7.5 mg gefapixant vs. placebo Week 6 estimated treatment differences (gefapixant vs. placebo) and corresponding 95% CIs were estimated using a MMRM model, which included fixed effects for treatment group, visit, country, treatment-by-visit interaction, and Baseline value as a covariate; Test type: Other; p = 0.1718, Mixed Effect Repeated Measures model; LS Mean Difference = -0.5, 95% CI 2-sided [-1.1 to 0.2]
Statistical Analysis 2: Comparison: Placebo vs Gefapixant 20 mg; Week 6 DCS Total Score: 20 mg gefapixant vs. placebo Week 6 estimated treatment differences (gefapixant vs. placebo) and corresponding 95% CIs were estimated using a MMRM model, which included fixed effects for treatment group, visit, country, treatment-by-visit interaction, and Baseline value as a covariate; Test type: Other; p = 0.0651, Mixed Effect Repeated Measures model; LS Mean Difference = -0.6, 95% CI 2-sided [-1.3 to 0.0]
Statistical Analysis 3: Comparison: Placebo vs Gefapixant 50 mg; Week 6 DCS Total Score: 50 mg gefapixant vs. placebo Week 6 estimated treatment differences (gefapixant vs. placebo) and corresponding 95% CIs were estimated using a MMRM model, which included fixed effects for treatment group, visit, country, treatment-by-visit interaction, and Baseline value as a covariate; Test type: Other; p = 0.0848, Mixed Effect Repeated Measures model; LS Mean Difference = -0.6, 95% CI 2-sided [-1.2 to 0.1]

41. Secondary Outcome: Change From Baseline in Weekly Mean DCS at Week 7
Description: as for outcome 35
Time Frame: Baseline, Week 7
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Gefapixant 7.5 mg | Gefapixant 20 mg | Gefapixant 50 mg
Number analyzed (Participants) | 61 | 59 | 59 | 57
score on a scale | -1.5 (0.25) | -1.7 (0.25) | -1.9 (0.25) | -1.9 (0.25)
Statistical Analysis 1: Comparison: Placebo vs Gefapixant 7.5 mg; Week 7 DCS Total Score: 7.5 mg gefapixant vs. placebo Week 7 estimated treatment differences (gefapixant vs. placebo) and corresponding 95% CIs were estimated using a MMRM model, which included fixed effects for treatment group, visit, country, treatment-by-visit interaction, and Baseline value as a covariate; Test type: Other; p = 0.6715, Mixed Effect Repeated Measures model; LS Mean Difference = -0.1, 95% CI 2-sided [-0.8 to 0.5]
Statistical Analysis 2: Comparison: Placebo vs Gefapixant 20 mg; Week 7 DCS Total Score: 20 mg gefapixant vs. placebo Week 7 estimated treatment differences (gefapixant vs. placebo) and corresponding 95% CIs were estimated using a MMRM model, which included fixed effects for treatment group, visit, country, treatment-by-visit interaction, and Baseline value as a covariate; Test type: Other; p = 0.3514, Mixed Effect Repeated Measures model; LS Mean Difference = -0.3, 95% CI 2-sided [-1.0 to 0.4]
Statistical Analysis 3: Comparison: Placebo vs Gefapixant 50 mg; Week 7 DCS Total Score: 50 mg gefapixant vs. placebo Week 7 estimated treatment differences (gefapixant vs. placebo) and corresponding 95% CIs were estimated using a MMRM model, which included fixed effects for treatment group, visit, country, treatment-by-visit interaction, and Baseline value as a covariate; Test type: Other; p = 0.2809, Mixed Effect Repeated Measures model; LS Mean Difference = -0.4, 95% CI 2-sided [-1.1 to 0.3]

42. Secondary Outcome: Change From Baseline in Weekly Mean DCS at Week 8
Description: as for outcome 35
Time Frame: Baseline, Week 8
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Gefapixant 7.5 mg | Gefapixant 20 mg | Gefapixant 50 mg
Number analyzed (Participants) | 61 | 59 | 59 | 57
score on a scale | -1.7 (0.25) | -1.8 (0.25) | -1.9 (0.25) | -1.9 (0.26)
Statistical Analysis 1: Comparison: Placebo vs Gefapixant 7.5 mg; Week 8 DCS Total Score: 7.5 mg gefapixant vs. placebo Week 8 estimated treatment differences (gefapixant vs. placebo) and corresponding 95% CIs were estimated using a MMRM model, which included fixed effects for treatment group, visit, country, treatment-by-visit interaction, and Baseline value as a covariate; Test type: Other; p = 0.6022, Mixed Effect Repeated Measures model; LS Mean Difference = -0.2, 95% CI 2-sided [-0.9 to 0.5]
Statistical Analysis 2: Comparison: Placebo vs Gefapixant 20 mg; Week 8 DCS Total Score: 20 mg gefapixant vs. placebo Week 8 estimated treatment differences (gefapixant vs. placebo) and corresponding 95% CIs were estimated using a MMRM model, which included fixed effects for treatment group, visit, country, treatment-by-visit interaction, and Baseline value as a covariate; Test type: Other; p = 0.4456, Mixed Effect Repeated Measures model; LS Mean Difference = -0.3, 95% CI 2-sided [-1.0 to 0.4]
Statistical Analysis 3: Comparison: Placebo vs Gefapixant 50 mg; Week 8 DCS Total Score: 50 mg gefapixant vs. placebo Week 8 estimated treatment differences (gefapixant vs. placebo) and corresponding 95% CIs were estimated using a MMRM model, which included fixed effects for treatment group, visit, country, treatment-by-visit interaction, and Baseline value as a covariate; Test type: Other; p = 0.4629, Mixed Effect Repeated Measures model; LS Mean Difference = -0.3, 95% CI 2-sided [-1.0 to 0.4]

43. Secondary Outcome: Change From Baseline in Weekly Mean DCS at Week 9
Description: as for outcome 35
Time Frame: Baseline, Week 9
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Gefapixant 7.5 mg | Gefapixant 20 mg | Gefapixant 50 mg
Number analyzed (Participants) | 61 | 59 | 59 | 57
score on a scale | -1.6 (0.25) | -1.9 (0.25) | -2.2 (0.25) | -2.0 (0.26)
Statistical Analysis 1: Comparison: Placebo vs Gefapixant 7.5 mg; Week 9 DCS Total Score: 7.5 mg gefapixant vs. placebo Week 9 estimated treatment differences (gefapixant vs. placebo) and corresponding 95% CIs were estimated using a MMRM model, which included fixed effects for treatment group, visit, country, treatment-by-visit interaction, and Baseline value as a covariate; Test type: Other; p = 0.3749, Mixed Effect Repeated Measures model; LS Mean Difference = -0.3, 95% CI 2-sided [-1.0 to 0.4]
Statistical Analysis 2: Comparison: Placebo vs Gefapixant 20 mg; Week 9 DCS Total Score: 20 mg gefapixant vs. placebo Week 9 estimated treatment differences (gefapixant vs. placebo) and corresponding 95% CIs were estimated using a MMRM model, which included fixed effects for treatment group, visit, country, treatment-by-visit interaction, and Baseline value as a covariate; Test type: Other; p = 0.0854, Mixed Effect Repeated Measures model; LS Mean Difference = -0.6, 95% CI 2-sided [-1.3 to 0.1]
Statistical Analysis 3: Comparison: Placebo vs Gefapixant 50 mg; Week 9 DCS Total Score: 50 mg gefapixant vs. placebo Week 9 estimated treatment differences (gefapixant vs. placebo) and corresponding 95% CIs were estimated using a MMRM model, which included fixed effects for treatment group, visit, country, treatment-by-visit interaction, and Baseline value as a covariate; Test type: Other; p = 0.2672, Mixed Effect Repeated Measures model; LS Mean Difference = -0.4, 95% CI 2-sided [-1.1 to 0.3]

44. Secondary Outcome: Change From Baseline in Weekly Mean DCS at Week 10
Description: as for outcome 35
Time Frame: Baseline, Week 10
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Gefapixant 7.5 mg | Gefapixant 20 mg | Gefapixant 50 mg
Number analyzed (Participants) | 61 | 59 | 59 | 57
score on a scale | -1.5 (0.25) | -1.6 (0.25) | -2.1 (0.25) | -2.1 (0.26)
Statistical Analysis 1: Comparison: Placebo vs Gefapixant 7.5 mg; Week 10 DCS Total Score: 7.5 mg gefapixant vs. placebo Week 10 estimated treatment differences (gefapixant vs. placebo) and corresponding 95% CIs were estimated using a MMRM model, which included fixed effects for treatment group, visit, country, treatment-by-visit interaction, and Baseline value as a covariate; Test type: Other; p = 0.7255, Mixed Effect Repeated Measures model; LS Mean Difference = -0.1, 95% CI 2-sided [-0.8 to 0.6]
Statistical Analysis 2: Comparison: Placebo vs Gefapixant 20 mg; Week 10 DCS Total Score: 20 mg gefapixant vs. placebo Week 10 estimated treatment differences (gefapixant vs. placebo) and corresponding 95% CIs were estimated using a MMRM model, which included fixed effects for treatment group, visit, country, treatment-by-visit interaction, and Baseline value as a covariate; Test type: Other; p = 0.0918, Mixed Effect Repeated Measures model; LS Mean Difference = -0.6, 95% CI 2-sided [-1.3 to 0.1]
Statistical Analysis 3: Comparison: Placebo vs Gefapixant 50 mg; Week 10 DCS Total Score: 50 mg gefapixant vs. placebo Week 10 estimated treatment differences (gefapixant vs. placebo) and corresponding 95% CIs were estimated using a MMRM model, which included fixed effects for treatment group, visit, country, treatment-by-visit interaction, and Baseline value as a covariate; Test type: Other; p = 0.1263, Mixed Effect Repeated Measures model; LS Mean Difference = -0.5, 95% CI 2-sided [-1.2 to 0.2]

45. Secondary Outcome: Change From Baseline in Weekly Mean DCS at Week 11
Description: as for outcome 35
Time Frame: Baseline, Week 11
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Gefapixant 7.5 mg | Gefapixant 20 mg | Gefapixant 50 mg
Number analyzed (Participants) | 61 | 59 | 59 | 57
score on a scale | -1.5 (0.25) | -1.8 (0.25) | -2.1 (0.25) | -2.2 (0.26)
Statistical Analysis 1: Comparison: Placebo vs Gefapixant 7.5 mg; Week 11 DCS Total Score: 7.5 mg gefapixant vs. placebo Week 11 estimated treatment differences (gefapixant vs. placebo) and corresponding 95% CIs were estimated using a MMRM model, which included fixed effects for treatment group, visit, country, treatment-by-visit interaction, and Baseline value as a covariate; Test type: Other; p = 0.4058, Mixed Effect Repeated Measures model; LS Mean Difference = -0.3, 95% CI 2-sided [-1.0 to 0.4]
Statistical Analysis 2: Comparison: Placebo vs Gefapixant 20 mg; Week 11 DCS Total Score: 20 mg gefapixant vs. placebo Week 11 estimated treatment differences (gefapixant vs. placebo) and corresponding 95% CIs were estimated using a MMRM model, which included fixed effects for treatment group, visit, country, treatment-by-visit interaction, and Baseline value as a covariate; Test type: Other; p = 0.0828, Mixed Effect Repeated Measures model; LS Mean Difference = -0.6, 95% CI 2-sided [-1.3 to 0.1]
Statistical Analysis 3: Comparison: Placebo vs Gefapixant 50 mg; Week 11 DCS Total Score: 50 mg gefapixant vs. placebo Week 11 estimated treatment differences (gefapixant vs. placebo) and corresponding 95% CIs were estimated using a MMRM model, which included fixed effects for treatment group, visit, country, treatment-by-visit interaction, and Baseline value as a covariate; Test type: Other; p = 0.0575, Mixed Effect Repeated Measures model; LS Mean Difference = -0.7, 95% CI 2-sided [-1.4 to 0.0]

46. Secondary Outcome: Change From Baseline in Weekly Mean DCS at Week 12
Description: as for outcome 35
Time Frame: Baseline, Week 12
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Gefapixant 7.5 mg | Gefapixant 20 mg | Gefapixant 50 mg
Number analyzed (Participants) | 61 | 59 | 59 | 57
score on a scale | -1.5 (0.26) | -1.8 (0.26) | -2.2 (0.26) | -2.2 (0.27)
Statistical Analysis 1: Comparison: Placebo vs Gefapixant 7.5 mg; Week 12 DCS Total Score: 7.5 mg gefapixant vs. placebo Week 12 estimated treatment differences (gefapixant vs. placebo) and corresponding 95% CIs were estimated using a MMRM model, which included fixed effects for treatment group, visit, country, treatment-by-visit interaction, and Baseline value as a covariate; Test type: Other; p = 0.4163, Mixed Effect Repeated Measures model; LS Mean Difference = -0.3, 95% CI 2-sided [-1.0 to 0.4]
Statistical Analysis 2: Comparison: Placebo vs Gefapixant 20 mg; Week 12 DCS Total Score: 20 mg gefapixant vs. placebo Week 12 estimated treatment differences (gefapixant vs. placebo) and corresponding 95% CIs were estimated using a MMRM model, which included fixed effects for treatment group, visit, country, treatment-by-visit interaction, and Baseline value as a covariate; Test type: Other; p = 0.0882, Mixed Effect Repeated Measures model; LS Mean Difference = -0.6, 95% CI 2-sided [-1.3 to 0.1]
Statistical Analysis 3: Comparison: Placebo vs Gefapixant 50 mg; Week 12 DCS Total Score: 50 mg gefapixant vs. placebo Week 12 estimated treatment differences (gefapixant vs. placebo) and corresponding 95% CIs were estimated using a MMRM model, which included fixed effects for treatment group, visit, country, treatment-by-visit interaction, and Baseline value as a covariate; Test type: Other; p = 0.0961, Mixed Effect Repeated Measures model; LS Mean Difference = -0.6, 95% CI 2-sided [-1.4 to 0.1]

47. Secondary Outcome: Change From Baseline in Leicester Cough Questionnaire (LCQ) Total Score After 4 Weeks of Treatment (Day 28)
Description: The LCQ instrument is designed to assess the impact of cough on various aspects of a participant's life over the preceding 2 weeks. It consists of 19 items which are divided over 3 domains: Physical (items 1, 2, 3, 9, 10, 11, 14 and 15), Psychological (4, 5, 6, 12, 13, 16, and 17), and Social (7, 8, 18, 19). A 7-point Likert scale is used to rate each item. For each domain, the domain score (range 1-7) is the sum of the individual item scores within the domain divided by the number of items in the domain. The total score is the sum of the three domain scores and ranges from 3-21; a higher score corresponds to a better health status. Baseline LCQ was defined as the LCQ collected at Baseline (Study Day -1). LS mean change from baseline in total LCQ score was reported for each treatment group with associated SE.
Time Frame: Baseline, Day 28
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Gefapixant 7.5 mg | Gefapixant 20 mg | Gefapixant 50 mg
Number analyzed (Participants) | 61 | 59 | 59 | 57
score on a scale | 2.1 (0.40) | 2.9 (0.40) | 2.3 (0.40) | 4.2 (0.4)
Statistical Analysis 1: Comparison: Placebo vs Gefapixant 7.5 mg; Day 28 LCQ Total Score: 7.5 mg gefapixant vs. placebo Day 28 estimated treatment differences (gefapixant vs. placebo) and corresponding 95% CIs were estimated using a MMRM model, which included fixed effects for treatment group, visit, country, treatment-by-visit interaction, and Baseline value as a covariate; Test type: Other; p = 0.1630, Mixed Effect Repeated Measures model; LS Mean Difference = 0.8, 95% CI 2-sided [-0.3 to 1.9]
Statistical Analysis 2: Comparison: Placebo vs Gefapixant 20 mg; Day 28 LCQ Total Score: 20 mg gefapixant vs. placebo Day 28 estimated treatment differences (gefapixant vs. placebo) and corresponding 95% CIs were estimated using a MMRM model, which included fixed effects for treatment group, visit, country, treatment-by-visit interaction, and Baseline value as a covariate; Test type: Other; p = 0.7601, Mixed Effect Repeated Measures model; LS Mean Difference = 0.2, 95% CI 2-sided [-1.0 to 1.3]
Statistical Analysis 3: Comparison: Placebo vs Gefapixant 50 mg; Day 28 LCQ Total Score: 50 mg gefapixant vs. placebo Day 28 estimated treatment differences (gefapixant vs. placebo) and corresponding 95% CIs were estimated using a MMRM model, which included fixed effects for treatment group, visit, country, treatment-by-visit interaction, and Baseline value as a covariate; Test type: Other; p = 0.0004, Mixed Effect Repeated Measures model; LS Mean Difference = 2.1, 95% CI 2-sided [0.9 to 3.2]

48. Secondary Outcome: Change From Baseline in Leicester Cough Questionnaire (LCQ) Total Score After 8 Weeks of Treatment (Day 56)
Description: as for outcome 47
Time Frame: Baseline, Day 56
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Gefapixant 7.5 mg | Gefapixant 20 mg | Gefapixant 50 mg
Number analyzed (Participants) | 61 | 59 | 59 | 57
score on a scale | 2.0 (0.4) | 3.1 (0.4) | 3.0 (0.4) | 3.5 (0.5)
Statistical Analysis 1: Comparison: Placebo vs Gefapixant 7.5 mg; Day 56 LCQ Total Score: 7.5 mg gefapixant vs. placebo Day 56 estimated treatment differences (gefapixant vs. placebo) and corresponding 95% CIs were estimated using a MMRM model, which included fixed effects for treatment group, visit, country, treatment-by-visit interaction, and Baseline value as a covariate; Test type: Other; p = 0.0941, Mixed Effect Repeated Measures model; LS Mean Difference = 1.0, 95% CI 2-sided [-0.2 to 2.3]
Statistical Analysis 2: Comparison: Placebo vs Gefapixant 20 mg; Day 56 LCQ Total Score: 20 mg gefapixant vs. placebo Day 56 estimated treatment differences (gefapixant vs. placebo) and corresponding 95% CIs were estimated using a MMRM model, which included fixed effects for treatment group, visit, country, treatment-by-visit interaction, and Baseline value as a covariate; Test type: Other; p = 0.1321, Mixed Effect Repeated Measures model; LS Mean Difference = 0.9, 95% CI 2-sided [-0.3 to 2.2]
Statistical Analysis 3: Comparison: Placebo vs Gefapixant 50 mg; Day 56 LCQ Total Score: 50 mg gefapixant vs. placebo Day 56 estimated treatment differences (gefapixant vs. placebo) and corresponding 95% CIs were estimated using a MMRM model, which included fixed effects for treatment group, visit, country, treatment-by-visit interaction, and Baseline value as a covariate; Test type: Other; p = 0.0192, Mixed Effect Repeated Measures model; LS Mean Difference = 1.5, 95% CI 2-sided [0.2 to 2.7]

49. Secondary Outcome: Change From Baseline in Leicester Cough Questionnaire (LCQ) Total Score At Day 85/Early Termination
Description: as for outcome 47
Time Frame: Baseline, Day 85/Early Termination
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Gefapixant 7.5 mg | Gefapixant 20 mg | Gefapixant 50 mg
Number analyzed (Participants) | 61 | 59 | 59 | 57
score on a scale | 2.1 (0.4) | 3.3 (0.4) | 3.2 (0.4) | 4.0 (0.5)
Statistical Analysis 1: Comparison: Placebo vs Gefapixant 7.5 mg; Day 85/Early Termination LCQ Total Score: 7.5 mg gefapixant vs. placebo Day 85/Early Termination estimated treatment differences (gefapixant vs. placebo) and corresponding 95% CIs were estimated using a MMRM model, which included fixed effects for treatment group, visit, country, treatment-by-visit interaction, and Baseline value as a covariate; Test type: Other; p = 0.0626, Mixed Effect Repeated Measures model; LS Mean Difference = 1.2, 95% CI 2-sided [-0.1 to 2.4]
Statistical Analysis 2: Comparison: Placebo vs Gefapixant 20 mg; Day 85/Early Termination LCQ Total Score: 20 mg gefapixant vs. placebo Day 85/Early Termination estimated treatment differences (gefapixant vs. placebo) and corresponding 95% CIs were estimated using a MMRM model, which included fixed effects for treatment group, visit, country, treatment-by-visit interaction, and Baseline value as a covariate; Test type: Other; p = 0.0967, Mixed Effect Repeated Measures model; LS Mean Difference = 1.0, 95% CI 2-sided [-0.2 to 2.3]
Statistical Analysis 3: Comparison: Placebo vs Gefapixant 50 mg; Day 85/Early Termination LCQ Total Score: 50 mg gefapixant vs. placebo Day 85/Early Termination estimated treatment differences (gefapixant vs. placebo) and corresponding 95% CIs were estimated using a MMRM model, which included fixed effects for treatment group, visit, country, treatment-by-visit interaction, and Baseline value as a covariate; Test type: Other; p = 0.0028, Mixed Effect Repeated Measures model; LS Mean Difference = 1.9, 95% CI 2-sided [0.7 to 3.1]

50. Secondary Outcome: Percentage of Participants Reporting "Very Much Improved" or "Much Improved" According to the Patient's Global Impression of Change (PGIC) After 4 Weeks of Treatment (Day 28)
Description: The self-reported measure Patient's Global Impression of Change (PGIC) reflects a participant's belief about the efficacy of treatment. PGIC is a 7-point scale depicting a patient's rating of overall improvement. Participants rate their change as "very much improved," "much improved," "minimally improved," "no change," "minimally worse," "much worse," or "very much worse." The counts and percentages of ordered responses to the participant's global perception of change were computed for each treatment group on Day 28 and the percentage of participants with improvements (either "very much improved" or "much improved" on the PGIC scale) was reported for each treatment group.
Time Frame: Day 28
Population: All randomized participants who had taken at least 1 dose of study medication and provided at least 1 baseline and 1 Day 28 PGIC observation during the treatment period.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Gefapixant 7.5 mg | Gefapixant 20 mg | Gefapixant 50 mg
Number analyzed (Participants) | 60 | 58 | 59 | 56
percentage of participants | 30.0 | 37.9 | 35.6 | 46.4
Statistical Analysis 1: Comparison: Placebo vs Gefapixant 7.5 mg; Day 28 PGIC: 7.5 mg gefapixant vs. placebo The distribution of responses were compared between each of the gefapixant treatment groups and placebo using the stratified CMH test (stratified by country). P-values calculated using CMH test; Test type: Superiority or Other; p = 0.3182, Cochran-Mantel-Haenszel
Statistical Analysis 2: Comparison: Placebo vs Gefapixant 20 mg; Day 28 PGIC: 20 mg gefapixant vs. placebo The distribution of responses were compared between each of the gefapixant treatment groups and placebo using the stratified CMH test (stratified by country). P-values calculated using CMH test; Test type: Superiority or Other; p = 0.5021, Cochran-Mantel-Haenszel
Statistical Analysis 3: Comparison: Placebo vs Gefapixant 50 mg; Day 28 PGIC: 50 mg gefapixant vs. placebo The distribution of responses were compared between each of the gefapixant treatment groups and placebo using the stratified CMH test (stratified by country). P-values calculated using CMH test; Test type: Superiority or Other; p = 0.0665, Cochran-Mantel-Haenszel

51. Secondary Outcome: Percentage of Participants Reporting "Very Much Improved" or "Much Improved" According to the PGIC After 8 Weeks of Treatment (Day 56)
Description: as for outcome 50
Time Frame: Day 56
Population: All randomized participants who had taken at least 1 dose of study medication and provided at least 1 baseline and 1 Day 56 PGIC observation during the treatment period.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Gefapixant 7.5 mg | Gefapixant 20 mg | Gefapixant 50 mg
Number analyzed (Participants) | 58 | 58 | 59 | 51
percentage of participants | 29.3 | 44.8 | 44.1 | 60.8
Statistical Analysis 1: Comparison: Placebo vs Gefapixant 7.5 mg; Day 56 PGIC: 7.5 mg gefapixant vs. placebo The distribution of responses were compared between each of the gefapixant treatment groups and placebo using the stratified CMH test (stratified by country). P-values calculated using CMH test; Test type: Superiority or Other; p = 0.0872, Cochran-Mantel-Haenszel
Statistical Analysis 2: Comparison: Placebo vs Gefapixant 20 mg; Day 56 PGIC: 20 mg gefapixant vs. placebo The distribution of responses were compared between each of the gefapixant treatment groups and placebo using the stratified CMH test (stratified by country). P-values calculated using CMH test; Test type: Superiority or Other; p = 0.0994, Cochran-Mantel-Haenszel
Statistical Analysis 3: Comparison: Placebo vs Gefapixant 50 mg; Day 56 PGIC: 50 mg gefapixant vs. placebo The distribution of responses were compared between each of the gefapixant treatment groups and placebo using the stratified CMH test (stratified by country). P-values calculated using CMH test; Test type: Superiority or Other; p = 0.0009, Cochran-Mantel-Haenszel

52. Secondary Outcome: Percentage of Participants Reporting "Very Much Improved" or "Much Improved" According to the PGIC at Day 85/Early Termination
Description: as for outcome 50
Time Frame: Day 85/Early Termination
Population: All randomized participants who had taken at least 1 dose of study medication and provided at least 1 baseline and 1 Day 85 PGIC observation during the treatment period.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Gefapixant 7.5 mg | Gefapixant 20 mg | Gefapixant 50 mg
Number analyzed (Participants) | 60 | 58 | 59 | 57
percentage of participants | 28.3 | 53.4 | 49.2 | 64.9
Statistical Analysis 1: Comparison: Placebo vs Gefapixant 7.5 mg; Day 85/Early Termination PGIC: 7.5 mg gefapixant vs. placebo The distribution of responses were compared between each of the gefapixant treatment groups and placebo using the stratified CMH test (stratified by country). P-values calculated using CMH test; Test type: Superiority or Other; p = 0.0037, Cochran-Mantel-Haenszel
Statistical Analysis 2: Comparison: Placebo vs Gefapixant 20 mg; Day 85/Early Termination PGIC: 20 mg gefapixant vs. placebo The distribution of responses were compared between each of the gefapixant treatment groups and placebo using the stratified CMH test (stratified by country). P-values calculated using CMH test; Test type: Superiority or Other; p = 0.0166, Cochran-Mantel-Haenszel
Statistical Analysis 3: Comparison: Placebo vs Gefapixant 50 mg; Day 85/Early Termination: 50 mg gefapixant vs. placebo The distribution of responses were compared between each of the gefapixant treatment groups and placebo using the stratified CMH test (stratified by country). P-values calculated using CMH test; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel

53. Secondary Outcome: Percentage of Participants Rated as "Very Much Improved" or "Much Improved" by Clinicians According to the Clinician's Global Impression of Change (CGIC) at Day 85/Early Termination
Description: The Clinician's Global Impression of Change (CGIC) reflects a clinician's belief about the efficacy of treatment. CGIC is a 7-point scale depicting a clinician's rating of a participant's overall improvement. Clinicians rated the participant's change at Week 12 (Day 85) as "very much improved," "much improved," "minimally improved," "no change," "minimally worse," "much worse," or "very much worse." The counts and percentages of ordered responses to the clinician's global perception of change were computed for each treatment group, and the percentage of participants rated by clinicians as having improvement (either "very much improved" or "much improved" on the CGIC scale) was reported for each treatment group.
Time Frame: Day 85/Early Termination
Population: All randomized participants who had taken at least 1 dose of study medication and provided at least 1 baseline and 1 Day 85 CGIC observation during the treatment period.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Gefapixant 7.5 mg | Gefapixant 20 mg | Gefapixant 50 mg
Number analyzed (Participants) | 60 | 58 | 59 | 57
percentage of participants | 35.0 | 53.4 | 50.8 | 64.9
Statistical Analysis 1: Comparison: Placebo vs Gefapixant 7.5 mg; Day 85/Early Termination CGIC: 7.5 mg gefapixant vs. placebo The distribution of responses were compared between each of the gefapixant treatment groups and placebo using the stratified CMH test (stratified by country). P-values calculated using CMH test; Test type: Superiority or Other; p = 0.0396, Cochran-Mantel-Haenszel
Statistical Analysis 2: Comparison: Placebo vs Gefapixant 20 mg; Day 85/Early Termination CGIC: 20 mg gefapixant vs. placebo The distribution of responses were compared between each of the gefapixant treatment groups and placebo using the stratified CMH test (stratified by country). P-values calculated using CMH test; Test type: Superiority or Other; p = 0.0751, Cochran-Mantel-Haenszel
Statistical Analysis 3: Comparison: Placebo vs Gefapixant 50 mg; Day 85/Early Termination CGIC: 50 mg gefapixant vs. placebo The distribution of responses were compared between each of the gefapixant treatment groups and placebo using the stratified CMH test (stratified by country). P-values calculated using CMH test; Test type: Superiority or Other; p = 0.0010, Cochran-Mantel-Haenszel

54. Secondary Outcome: Acceptability Questionnaire: Percentage of Participants That Were Likely to Take Study Medication For At Least One Year
Description: At the end of the treatment period (Day 85), participants were asked "How likely would you be to take this medication?" This question was asked in reference to the time frame of "At least one year". The counts and percentages of ordered categorical responses to this question were computed for each treatment group.
Time Frame: Day 85/Early Termination
Population: All randomized participants who had taken at least 1 dose of study medication and had available Acceptability Questionnaire data for the one year question at Day 85.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Gefapixant 7.5 mg | Gefapixant 20 mg | Gefapixant 50 mg
Number analyzed (Participants) | 60 | 58 | 58 | 57
percentage of participants
  Extremely unlikely | 3.3 | 6.9 | 5.2 | 1.8
  Unlikely | 3.3 | 1.7 | 3.4 | 12.3
  Neither likely or unlikely | 5.0 | 5.2 | 12.1 | 1.8
  Likely | 30.0 | 15.5 | 13.8 | 29.8
  Extremely likely | 58.3 | 70.7 | 65.5 | 54.4
Statistical Analysis 1: Comparison: Placebo vs Gefapixant 7.5 mg; 1 Year Acceptability: 7.5 mg gefapixant vs. placebo The distribution of "Extremely likely" responses was compared between each of the gefapixant treatment groups and placebo using the stratified CMH test (stratified by country). P-values calculated for the gefapixant vs. placebo using CMH test; Test type: Superiority or Other; p = 0.8464, Cochran-Mantel-Haenszel
Statistical Analysis 2: Comparison: Placebo vs Gefapixant 20 mg; 1 Year Acceptability: 20 mg gefapixant vs. placebo The distribution of "Extremely likely" responses was compared between each of the gefapixant treatment groups and placebo using the stratified CMH test (stratified by country). P-values calculated for gefapixant vs. placebo using CMH test; Test type: Superiority or Other; p = 0.7687, Cochran-Mantel-Haenszel
Statistical Analysis 3: Comparison: Placebo vs Gefapixant 50 mg; 1 Year Acceptability: 50 mg gefapixant vs. placebo The distribution of "Extremely likely" responses was compared between each of the gefapixant treatment groups and placebo using the stratified CMH test (stratified by country). P-values calculated for gefapixant vs. placebo using CMH test; Test type: Superiority or Other; p = 0.4364, Cochran-Mantel-Haenszel

55. Secondary Outcome: Acceptability Questionnaire: Percentage of Participants That Were Likely to Take Study Medication For At Least Six Months
Description: At the end of the treatment period (Day 85), participants were asked "How likely would you be to take this medication?" This question was asked in reference to the time frame of "At least six months". The counts and percentages of ordered categorical responses to this question were computed for each treatment group.
Time Frame: Day 85/Early Termination
Population: All randomized participants who had taken at least 1 dose of study medication and had available Acceptability Questionnaire data for the six month question at Day 85.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Gefapixant 7.5 mg | Gefapixant 20 mg | Gefapixant 50 mg
Number analyzed (Participants) | 60 | 57 | 58 | 57
percentage of participants
  Extremely unlikely | 3.3 | 5.3 | 5.2 | 1.8
  Unlikely | 1.7 | 3.5 | 3.4 | 10.5
  Neither likely or unlikely | 6.7 | 3.5 | 6.9 | 3.5
  Likely | 21.7 | 14.0 | 17.2 | 29.8
  Extremely likely | 66.7 | 73.7 | 67.2 | 54.4
Statistical Analysis 1: Comparison: Placebo vs Gefapixant 7.5 mg; 6 Month Acceptability: 7.5 mg gefapixant vs. placebo The distribution of "Extremely likely" responses were compared between each of the gefapixant treatment groups and placebo using the stratified CMH test (stratified by country). P-values calculated for gefapixant vs. placebo using CMH test; Test type: Superiority or Other; p = 0.9966, Cochran-Mantel-Haenszel
Statistical Analysis 2: Comparison: Placebo vs Gefapixant 20 mg; 6 Month Acceptability: 20 mg gefapixant vs. placebo The distribution of "Extremely likely" responses were compared between each of the gefapixant treatment groups and placebo using the stratified CMH test (stratified by country). P-values calculated for gefapixant vs. placebo using CMH test; Test type: Superiority or Other; p = 0.6372, Cochran-Mantel-Haenszel
Statistical Analysis 3: Comparison: Placebo vs Gefapixant 50 mg; 6 Month Acceptability: 50 mg gefapixant vs. placebo The distribution of "Extremely likely" responses were compared between each of the gefapixant treatment groups and placebo using the stratified CMH test (stratified by country). P-values calculated for gefapixant vs. placebo using CMH test; Test type: Superiority or Other; p = 0.2155, Cochran-Mantel-Haenszel

56. Secondary Outcome: Acceptability Questionnaire: Percentage of Participants That Were Likely to Take Study Medication For At Least Four Weeks
Description: At the end of the treatment period (Day 85), participants were asked "How likely would you be to take this medication?" This question was asked in reference to the time frame of "At least four weeks". The counts and percentages of ordered categorical responses to this question were computed for each treatment group.
Time Frame: Day 85/Early Termination
Population: All randomized participants who had taken at least 1 dose of study medication and had available Acceptability Questionnaire data for the four week question at Day 85.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Gefapixant 7.5 mg | Gefapixant 20 mg | Gefapixant 50 mg
Number analyzed (Participants) | 60 | 58 | 58 | 57
percentage of participants
  Extremely unlikely | 3.3 | 5.2 | 5.2 | 0.0
  Unlikely | 1.7 | 1.7 | 1.7 | 5.3
  Neither likely or unlikely | 3.3 | 1.7 | 6.9 | 8.8
  Likely | 18.3 | 19.0 | 15.5 | 26.3
  Extremely likely | 73.3 | 72.4 | 70.7 | 59.6
Statistical Analysis 1: Comparison: Placebo vs Gefapixant 7.5 mg; 4 Week Acceptability: 7.5 mg gefapixant vs. placebo The distribution of "Extremely likely" responses were compared between each of the gefapixant treatment groups and placebo using the stratified CMH test (stratified by country). P-values calculated for gefapixant vs. placebo using CMH test; Test type: Superiority or Other; p = 0.7559, Cochran-Mantel-Haenszel
Statistical Analysis 2: Comparison: Placebo vs Gefapixant 20 mg; 4 Week Acceptability: 20 mg gefapixant vs. placebo The distribution of "Extremely likely" responses were compared between each of the gefapixant treatment groups and placebo using the stratified CMH test (stratified by country). P-values calculated for gefapixant vs. placebo using CMH test; Test type: Superiority or Other; p = 0.5091, Cochran-Mantel-Haenszel
Statistical Analysis 3: Comparison: Placebo vs Gefapixant 50 mg; 4 Week Acceptability: 50 mg gefapixant vs. placebo The distribution of "Extremely likely" responses were compared between each of the gefapixant treatment groups and placebo using the stratified CMH test (stratified by country). P-values calculated for gefapixant vs. placebo using CMH test; Test type: Superiority or Other; p = 0.2790, Cochran-Mantel-Haenszel

57. Secondary Outcome: Acceptability Questionnaire: Percentage of Participants That Were Likely to Take Study Medication Twice Daily
Description: At the end of the treatment period (Day 85), participants were asked "How likely would you be to take this medication?" This question was asked in reference to the time frame of "Twice daily". The counts and percentages of ordered categorical responses to this question were computed for each treatment group.
Time Frame: Day 85/Early Termination
Population: All randomized participants who had taken at least 1 dose of study medication and had available Acceptability Questionnaire data for the twice daily question at Day 85.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Gefapixant 7.5 mg | Gefapixant 20 mg | Gefapixant 50 mg
Number analyzed (Participants) | 60 | 57 | 57 | 56
percentage of participants
  Extremely unlikely | 3.3 | 7.0 | 5.3 | 1.8
  Unlikely | 0.0 | 0.0 | 3.5 | 5.4
  Neither likely or unlikely | 3.3 | 5.3 | 3.5 | 8.9
  Likely | 20.0 | 15.8 | 22.8 | 30.4
  Extremely likely | 73.3 | 71.9 | 64.9 | 53.6
Statistical Analysis 1: Comparison: Placebo vs Gefapixant 7.5 mg; Twice Daily Acceptability: 7.5 mg gefapixant vs. placebo The distribution of "Extremely likely" responses were compared between each of the gefapixant treatment groups and placebo using the stratified CMH test (stratified by country). P-values calculated for gefapixant vs. placebo using CMH test; Test type: Superiority or Other; p = 0.3887, Cochran-Mantel-Haenszel
Statistical Analysis 2: Comparison: Placebo vs Gefapixant 20 mg; Twice Daily Acceptability: 20 mg gefapixant vs. placebo The distribution of "Extremely likely" responses were compared between each of the gefapixant treatment groups and placebo using the stratified CMH test (stratified by country). P-values calculated for gefapixant vs. placebo using CMH test; Test type: Superiority or Other; p = 0.2333, Cochran-Mantel-Haenszel
Statistical Analysis 3: Comparison: Placebo vs Gefapixant 50 mg; Twice Daily Acceptability: 50 mg gefapixant vs. placebo The distribution of "Extremely likely" responses were compared between each of the gefapixant treatment groups and placebo using the stratified CMH test (stratified by country). P-values calculated for gefapixant vs. placebo using CMH test; Test type: Superiority or Other; p = 0.0534, Cochran-Mantel-Haenszel

58. Secondary Outcome: Taste Questionnaire: Percentage of Participants That Experienced Taste Effect After Taking Medication by Frequency After 12 Weeks of Treatment (Day 84)
Description: The tolerance to taste-related adverse events (AEs) was evaluated at the end of the study (Day 84) and a structured taste questionnaire was administered to participants experiencing a taste-related AE. Participants were asked to indicate the frequency that they experienced the taste effect by answering the question "How frequently do you experience the taste effect after taking each dose of medication?" The counts and percentages of categorical frequency responses to the individual items were computed for each treatment group.
Time Frame: Day 84
Population: All randomized participants who had taken at least 1 dose of study medication, who had experienced a taste-related AE, and who had Day 84 taste questionnaire data available.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Gefapixant 7.5 mg | Gefapixant 20 mg | Gefapixant 50 mg
Number analyzed (Participants) | 57 | 56 | 57 | 51
percentage of participants
  No Taste Effect Noted | 96.5 | 96.4 | 61.4 | 35.3
  Never | 1.8 | 0.0 | 0.0 | 0.0
  Occasionally | 1.8 | 1.8 | 8.8 | 0.0
  Often | 0.0 | 1.8 | 7.0 | 3.9
  Almost Always | 0.0 | 0.0 | 7.0 | 9.8
  Always | 0.0 | 0.0 | 15.8 | 51.0
  No Taste Effect Noted + Never | 98.2 | 96.4 | 61.4 | 35.3
Statistical Analysis 1: Comparison: Placebo vs Gefapixant 7.5 mg; Taste Effect Frequency: 7.5 mg gefapixant vs. placebo The distribution of "No Taste Effect Noted" or "Never" responses were compared between each of the gefapixant treatment groups and placebo using the stratified CMH test (stratified by country). P-values calculated for gefapixant vs. placebo using CMH test; Test type: Superiority or Other; p = 0.6115, Cochran-Mantel-Haenszel
Statistical Analysis 2: Comparison: Placebo vs Gefapixant 20 mg; Taste Effect Frequency: 20 mg gefapixant vs. placebo The distribution of "No Taste Effect Noted" or "Never" responses were compared between each of the gefapixant treatment groups and placebo using the stratified CMH test (stratified by country). P-values calculated for gefapixant vs. placebo using CMH test; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel
Statistical Analysis 3: Comparison: Placebo vs Gefapixant 50 mg; Taste Effect Frequency: 50 mg gefapixant vs. placebo The distribution of "No Taste Effect Noted" or "Never" responses were compared between each of the gefapixant treatment groups and placebo using the stratified CMH test (stratified by country). P-values calculated for gefapixant vs. placebo using CMH test; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel

59. Secondary Outcome: Taste Questionnaire: Percentage of Participants That Found Taste Effect of Study Medication Bothersome After 12 Weeks of Treatment (Day 84)
Description: The tolerance to taste-related adverse events (AEs) was evaluated at the end of the study (Day 84) and a structured taste questionnaire was administered to participants experiencing a taste-related AE to determine what degree the participant found the taste effect bothersome by answering the question "How bothersome is the taste effect of the medication? The counts and percentages of categorical responses to the individual items were computed for each treatment group.
Time Frame: Day 84
Population: as for outcome 58
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Gefapixant 7.5 mg | Gefapixant 20 mg | Gefapixant 50 mg
Number analyzed (Participants) | 57 | 56 | 57 | 51
percentage of participants
  No Taste Effect Noted | 96.5 | 96.4 | 61.4 | 35.3
  Not At All | 3.5 | 3.6 | 7.0 | 5.9
  A Little | 0.0 | 0.0 | 8.8 | 3.9
  Somewhat | 0.0 | 0.0 | 17.5 | 13.7
  Very | 0.0 | 0.0 | 5.3 | 29.4
  Extremely | 0.0 | 0.0 | 0.0 | 11.8
  No Taste Effect Noted + Not At All | 100.0 | 100.0 | 68.4 | 41.2
Statistical Analysis 1: Comparison: Placebo vs Gefapixant 7.5 mg; Taste Effect Frequency: 7.5 mg gefapixant vs. placebo The distribution of "No Taste Effect Noted" or "Not at All" responses were compared between each of the gefapixant treatment groups and placebo using the stratified CMH test (stratified by country). P-values calculated for gefapixant vs. placebo using CMH test; Test type: Superiority or Other; p = 0, Cochran-Mantel-Haenszel — A p-value of zero was calculated if all participants (100%) had "No Taste Effect Noted" or "Not at All" responses in both comparison groups
Statistical Analysis 2: Comparison: Placebo vs Gefapixant 20 mg; Taste Effect Frequency: 20 mg gefapixant vs. placebo The distribution of "No Taste Effect Noted" or "Not at All" responses were compared between each of the gefapixant treatment groups and placebo using the stratified CMH test (stratified by country). P-values calculated for gefapixant vs. placebo using CMH test; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel
Statistical Analysis 3: Comparison: Placebo vs Gefapixant 50 mg; Taste Effect Frequency: 50 mg gefapixant vs. placebo The distribution of "No Taste Effect Noted" or "Not at All" responses were compared between each of the gefapixant treatment groups and placebo using the stratified CMH test (stratified by country). P-values calculated for gefapixant vs. placebo using CMH test; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel

ADVERSE EVENTS:
Time Frame: Up to ~14 weeks (Day 99)
Description: All randomized participants who received at least 1 dose of study drug. One participant randomized to receive 7.5 mg gefapixant was discontinued before receiving treatment.
Arm/Group | Placebo | Gefapixant 7.5 mg | Gefapixant 20 mg | Gefapixant 50 mg
Serious Adverse Events (participants affected / at risk) | 0/63 | 0/63 | 0/63 | 1/63
Other Adverse Events (participants affected / at risk) | 21/63 | 26/63 | 45/63 | 52/63
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=63) | Gefapixant 7.5 mg (N=63) | Gefapixant 20 mg (N=63) | Gefapixant 50 mg (N=63)
Frostbite (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=63) | Gefapixant 7.5 mg (N=63) | Gefapixant 20 mg (N=63) | Gefapixant 50 mg (N=63)
Dry mouth (Gastrointestinal disorders) | 6 (7) | 2 (2) | 3 (3) | 3 (3)
Hypoaesthesia oral (Gastrointestinal disorders) | 3 (4) | 2 (2) | 4 (4) | 5 (5)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 4 (4) | 6 (6)
Paraesthesia oral (Gastrointestinal disorders) | 5 (8) | 4 (6) | 5 (5) | 4 (4)
Nasopharyngitis (Infections and infestations) | 2 (3) | 0 (0) | 4 (4) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 2 (2) | 5 (5) | 9 (9) | 6 (6)
Urinary tract infection (Infections and infestations) | 2 (2) | 3 (3) | 5 (6) | 2 (3)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 5 (5) | 2 (2) | 0 (0)
Ageusia (Nervous system disorders) | 1 (1) | 0 (0) | 3 (3) | 13 (14)
Dysgeusia (Nervous system disorders) | 3 (4) | 6 (7) | 21 (26) | 30 (39)
Headache (Nervous system disorders) | 3 (4) | 4 (4) | 12 (16) | 4 (4)
Hypogeusia (Nervous system disorders) | 1 (1) | 0 (0) | 11 (12) | 15 (18)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (3) | 5 (5) | 5 (5)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 0 (0) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
In order to ensure that the Sponsor will be able to make comments and suggestions where pertinent, material for public dissemination will be submitted to the Sponsor for review at least sixty (60) days prior to submission for publication, public dissemination, or review by a publication committee. All reasonable comments made by the Sponsor in relation to a proposed publication by the Trust, University and/or the Investigator will be incorporated into the publication.